CLINICAL TRIAL: NCT03760029
Title: A NATURAL HISTORY STUDY IN CHINESE MALE PATIENTS WITH DUCHENNE MUSCULAR DYSTROPHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C3391004
Record Dates: First submitted 2018-11-15; First posted 2018-11-30 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Other): All subjects in this study will be observed for 24-30 months.
  Interventions: Other: Visit frequency

INTERVENTIONS:
Other: Visit frequency — All subjects need to visit sites more frequently than in routine clinical practice.

SUMMARY:
This is a multicenter, prospective, single cohort study designed to describe the natural history of DMD in Chinese male patients. A total of approximately 330 subjects will be enrolled with the target number of subjects in each group as below:

* Group 1, Ambulatory subjects aged <6 years, approximately 100 subjects;
* Group 2, Ambulatory subjects aged >=6 years, approximately 180 subjects;
* Group 3, Non-ambulatory subjects, approximately 50 subjects. Subjects will visit sites every 6 months. Each subject will be observed for at least 24 months. All subjects will remain enrolled until the study completion date, such that some will have data collected after Month 24. Subjects, who complete Visit 5/Month 24 at least 6 months prior to study completion, will be asked to complete an additional visit at Month 30.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male patients with any age, diagnosed with DMD. Diagnosis must be confirmed in subject's medical history and by genetic testing obtained during routine clinical care for diagnostic purposes as reported from an appropriate regulated laboratory using a clinically validated genetic test (genetic testing is not provided by the sponsor).
2. Subjects who are >=4 years old must be receiving glucocorticosteroids for a minimum of 6 months prior to signing informed consent. There should be no significant change (<0.2 mg/kg) in dosage or dose regimen (not related to body weight change) for at least 3 months immediately prior to signing the informed consent. Subjects who are aged >4 years will be exempt from this requirement; those not taking GC will be eligible if the initiation of GC treatment in these subjects is considered inappropriate in the opinion of Investigators.

Exclusion Criteria:

1. Any injury which may impact functional testing. Previous injuries must be fully healed prior to consenting. Prior lower limb fractures must be fully healed and at least 3 months from injury date.
2. Presence or history of other musculoskeletal or neurologic disease or somatic disorder not related to DMD including pulmonary, cardiac, and cognitive diseases.
3. Subjects >=4 years old who have not completed the varicella vaccination.
4. Participation in other studies involving investigational drug(s) for a minimum of 90 days prior to signing the informed consent and/or during study participation.

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 312 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- China (8):
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Children's Hospital of Chongqing Medical University (Liangjiang Branch), Chongqing, Chongqing Municipality
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou, Fujian
  - Peking University First Hospital, Beijing
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Huashan Hospital, Fudan University, Shanghai
  - Affiliated children's hospital of fudan university, Shanghai
  - Children's Hospital of Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Li X, Lv J, Zhu W, Hong S, Wang Z, Chang X, Gao YX, Zhou Y, Jia C, Fang J, Patterson TA. A 1-year analysis from a natural history study in Chinese individuals with Duchenne muscular dystrophy. Lancet Reg Health West Pac. 2023 Nov 28;42:100944. doi: 10.1016/j.lanwpc.2023.100944. eCollection 2024 Jan. PMID 38089167
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3391004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, prospective study to describe natural history of Duchenne muscular dystrophy (DMD) in Chinese male participants.
Pre-assignment Details: A total of 318 participants were screened of which 6 were screen failures and 312 participants were enrolled at 6 sites in China.
Groups:
- Ambulatory Participants With Age <6 Years: Participants diagnosed with DMD who were ambulant and were less than 6 years of age at the time of screening were included. No investigational drug was administered, and participants were allowed to take medications prescribed by their physicians, which constituted the standard of care (SOC).
- Ambulatory Participants With Age >=6 Years: Participants diagnosed with DMD who were ambulant and were greater than or equal to (>=6) years of age at the time of screening were included. No investigational drug was administered, and participants were allowed to take medications prescribed by their physicians, which constituted the SOC.
- Non-ambulatory Participants: Participants diagnosed with DMD who were non-ambulatory (i.e., used wheel chair full-time or were unable to complete daily activities [such as going to bathroom] by walking independently, based on performance reported at home by participant or caregiver and verification by trained clinical evaluator [CE] with the inability to perform the 10-meter run/walk assessment) were included. No investigational drug was administered, and participants were allowed to take medications prescribed by their physicians, which constituted the SOC.
Period: Overall Study
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants
Started | 99 | 177 | 36
Completed | 91 | 166 | 33
Not Completed | 8 | 11 | 3
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 4 | 1
Not completed — Withdrawal by parent/guardian | 4 | 4 | 1
Not completed — Other | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all participants who had been enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total
Number analyzed (Participants) | 99 | 177 | 36 | 312
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.0 (1.23) | 9.0 (1.99) | 12.7 (2.71) | 7.9 (3.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 99 | 177 | 36 | 312
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 99 | 177 | 36 | 312
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 99 | 177 | 36 | 312
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Age of Participants When They Failed to Walk
Description: Participant's age at life-altering clinical milestones- failure to walk was calculated based on the birthdate and the date of failure to walk as reported by caregiver during 30 months of this study. Participants who were not reported being failure to walk by their caregivers were censored on the day of their last visit. Kaplan-Meier method was used for analysis.
Time Frame: Up to Month 30
Population: Full Analysis Set included all participants who had been enrolled in the study. Here, 'Number of Participants Analyzed' signifies participants included in the Kaplan-Meier analysis. No participant in "Ambulatory participants aged < 6 years" had an event of "failure to walk".
Measure: Median (95% Confidence Interval); unit: Years
Groups:
- Total Ambulatory Participants: Participants diagnosed with DMD who were ambulant at the time of screening were included. No investigational drug was administered, and participants were allowed to take medications prescribed by their physicians, which constituted the SOC.
- Total Participants: Participants diagnosed with DMD who were ambulant and who were non-ambulatory (i.e., used wheel chair full-time or were unable to complete daily activities [such as going to bathroom] by walking independently, based on performance reported at home by participant or caregiver and verification by trained CE with the inability to perform the 10-meter run/walk assessment) were included.
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 177 | 276 | 36 | 312
Years | NA [NA to NA] — Data could not be estimated as no participants had "failure to walk" event | 14.4 [13.9 to NA] — The upper limit of the 95% confidence interval was not reached due to less number of participants with an event. | 14.4 [13.9 to NA] — The upper limit of the 95% confidence interval was not reached due to less number of participants with an event. | 11.1 [10.0 to 11.4] | 13.1 [12.5 to 14.1]

2. Primary Outcome: Age of Participants When They Failed to Stand
Description: Participant's age at life-altering clinical milestones- failure to stand was calculated based on the birthdate and the date of failure to stand as reported by caregiver during 30 months of this study. Participants who were not reported being failure to stand by their caregivers were censored on the day of their last visit. Kaplan-Meier method was used for analysis.
Time Frame: Up to Month 30
Population: Full Analysis Set included all participants who had been enrolled in the study. Here, 'Number of Participants Analyzed' signifies participants included in the Kaplan-Meier analysis. No participant in "Ambulatory participants aged <6 years" had an event of "failure to stand".
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 177 | 276 | 36 | 312
Years | NA [NA to NA] — Data could not be estimated as no participants had "failure to stand" event | 14.4 [13.9 to NA] — The upper limit of the 95% confidence interval was not reached due to less number of participants with an event. | 14.4 [13.9 to NA] — The upper limit of the 95% confidence interval was not reached due to less number of participants with an event. | 11.0 [10.5 to 11.5] | 13.1 [12.9 to 14.4]

3. Primary Outcome: Age of Participants When They Failed to Self-feed
Description: Participant's age at life-altering clinical milestones- failure to self-feed during 30 months of this study was analyzed using the Kaplan-Meier method. Age was summarized in years.
Time Frame: Up to Month 30
Population: Full Analysis Set included all participants who had been enrolled in the study. Here, 'Number of Participants Analyzed' signifies participants included in the Kaplan-Meier analysis. No participant in "Ambulatory participants aged <6 years and >=6 years" had an event of "failure to self-feed".
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 177 | 276 | 36 | 312
Years | NA [NA to NA] — Data could not be estimated as no participants had "failure to self-feed" event | NA [NA to NA] — Data could not be estimated as no participants had "failure to self-feed" event | NA [NA to NA] — Data could not be estimated as no participants had "failure to self-feed" event | 20.0 [17.0 to NA] — The upper limit of the 95% confidence interval was not reached due to less number of participants with an event. | 20.0 [17.0 to NA] — The upper limit of the 95% confidence interval was not reached due to less number of participants with an event.

4. Primary Outcome: Change From Baseline in Northstar Ambulatory Assessment (NSAA) Total Score at Month 6: Ambulatory Participants Aged >=3 Years
Description: NSAA is a 17-item test that grades performance of various functional skills using the following scale: 0 (unable to achieve goal independently), 1 (modified method but achieves goal with no physical assistance), or 2 ("normal"- no obvious modification of activity). The scale assesses activities required to remain functionally ambulant (e.g. rise from the floor), activities that can be difficult even early in the disease (example [e.g.] standing on heels) and activities that are known to progressively deteriorate over time (stand from a chair, walk). NSAA total score was calculated by adding the responses of all 17 items and ranged from 0 to 34, with higher scores indicating better function. NSAA was only performed in ambulatory participants aged >=3 years old as pre-specified in protocol.
Time Frame: Baseline (Day 1) and Month 6
Population: Full Analysis Set included all participants who had been enrolled in the study. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants
Number analyzed (Participants) | 64 | 154 | 218
Units on a scale | 1.3 (4.44) | -1.0 (3.98) | -0.3 (4.24)

5. Primary Outcome: Change From Baseline in NSAA Total Score at Month 12: Ambulatory Participants Aged >=3 Years
Description: NSAA is a 17-item test that grades performance of various functional skills using the following scale: 0 (unable to achieve goal independently), 1 (modified method but achieves goal with no physical assistance), or 2 ("normal"- no obvious modification of activity). The scale assesses activities required to remain functionally ambulant (e.g. rise from the floor), activities that can be difficult even early in the disease (e.g. standing on heels) and activities that are known to progressively deteriorate over time (stand from a chair, walk). NSAA total score was calculated by adding the responses of all 17 items and ranged from 0 to 34, with higher scores indicating better function. NSAA was only performed in ambulatory participants aged >=3 years old as pre-specified in protocol.
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Ambulatory Participants: Participants diagnosed with DMD who were ambulant at the time of screening were included. No investigational drug was administered, and participants were allowed to take medications prescribed by their physicians, which constituted the SOC.
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Ambulatory Participants
Number analyzed (Participants) | 51 | 145 | 196
Units on a scale | 2.7 (5.37) | -2.1 (4.88) | -0.9 (5.42)

6. Primary Outcome: Change From Baseline in NSAA Total Score at Month 18: Ambulatory Participants Aged >=3 Years
Description: as for outcome 5
Time Frame: Baseline (Day 1) and Month 18
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants
Number analyzed (Participants) | 47 | 103 | 150
Units on a scale | 4.1 (5.12) | -3.6 (4.53) | -1.2 (5.93)

7. Primary Outcome: Change From Baseline in NSAA Total Score at Month 24: Ambulatory Participants Aged >=3 Years
Description: as for outcome 5
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants
Number analyzed (Participants) | 53 | 114 | 167
Units on a scale | 3.9 (4.67) | -4.9 (5.22) | -2.1 (6.50)

8. Primary Outcome: Change From Baseline in NSAA Total Score at Month 30: Ambulatory Participants Aged >=3 Years
Description: as for outcome 5
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants
Number analyzed (Participants) | 19 | 66 | 85
Units on a scale | 4.1 (5.09) | -5.9 (5.56) | -3.6 (6.84)

9. Primary Outcome: Change From Baseline in Performance of Upper Limb (PUL) 2.0 Total Score at Month 6: Participants Aged >=10 Years
Description: PUL 2.0 scale is a 22-item scale used to assess the change that occurs in motor performance of the upper limb overtime from when a participant is still ambulant to the time participant loses all arm function when non-ambulant. PUL 2.0 includes an entry item to define broad starting functional level and 22 items subdivided into shoulder level (six items), mid-level (nine items), and distal level (seven items). Each dimension (shoulder, mid, distal) can be scored separately. There is maximum score of 12 for shoulder level, 17 for mid-level, and 13 for distal level. The total score was calculated by adding three level scores and ranged from 0-42. Higher score indicates better upper limb function. PUL 2.0 total score was assessed in participants aged >=10 years only as pre-specified in protocol.
Time Frame: Baseline (Day 1) and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 46 | 4 | 50
Units on a scale | -0.0 (2.33) | -0.8 (2.22) | -0.1 (2.31)

10. Primary Outcome: Change From Baseline in PUL 2.0 Total Score at Month 12: Participants Aged >=10 Years
Description: as for outcome 9
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 43 | 23 | 66
Units on a scale | -0.6 (2.16) | -0.9 (2.37) | -0.7 (2.22)

11. Primary Outcome: Change From Baseline in PUL 2.0 Total Score at Month 18: Participants Aged >=10 Years
Description: as for outcome 9
Time Frame: Baseline (Day 1) and Month 18
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 27 | 4 | 31
Units on a scale | -1.7 (3.22) | -4.3 (2.75) | -2.1 (3.23)

12. Primary Outcome: Change From Baseline in PUL 2.0 Total Score at Month 24: Participants Aged >=10 Years
Description: as for outcome 9
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 35 | 21 | 56
Units on a scale | -2.8 (3.92) | -2.9 (3.23) | -2.8 (3.65)

13. Primary Outcome: Change From Baseline in PUL 2.0 Total Score at Month 30: Participants Aged >=10 Years
Description: as for outcome 9
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 18 | 4 | 22
Units on a scale | -1.7 (3.37) | -3.8 (1.71) | -2.1 (3.21)

14. Primary Outcome: Change From Baseline in Rise From Floor Velocity at Month 6: Ambulatory Participants Aged >=3 Years Only
Description: The rise from floor velocity was defined as the reciprocal of the time (in seconds) to rise from floor. The rise from floor test was performed only in ambulatory participants aged >=3 years old as pre-specified in the protocol.
Time Frame: Baseline (Day 1) and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Rise per second
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants
Number analyzed (Participants) | 75 | 155 | 230
Rise per second | 0.0 (0.07) | -0.0 (0.05) | 0.0 (0.06)

15. Primary Outcome: Change From Baseline in Rise From Floor Velocity at Month 12: Ambulatory Participants Aged >=3 Years Only
Description: as for outcome 14
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Rise per second
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants
Number analyzed (Participants) | 60 | 145 | 205
Rise per second | 0.0 (0.08) | -0.0 (0.07) | -0.0 (0.08)

16. Primary Outcome: Change From Baseline in Rise From Floor Velocity at Month 18: Ambulatory Participants Aged >=3 Years Only
Description: as for outcome 14
Time Frame: Baseline (Day 1) and Month 18
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Rise per second
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants
Number analyzed (Participants) | 57 | 104 | 161
Rise per second | 0.0 (0.08) | -0.0 (0.06) | -0.0 (0.08)

17. Primary Outcome: Change From Baseline in Rise From Floor Velocity at Month 24: Ambulatory Participants Aged >=3 Years Only
Description: as for outcome 14
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Rise per second
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants
Number analyzed (Participants) | 61 | 115 | 176
Rise per second | 0.0 (0.09) | -0.1 (0.07) | -0.0 (0.09)

18. Primary Outcome: Change From Baseline in Rise From Floor Velocity at Month 30: Ambulatory Participants Aged >=3 Years Only
Description: as for outcome 14
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Rise per second
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants
Number analyzed (Participants) | 22 | 67 | 89
Rise per second | 0.0 (0.10) | -0.1 (0.08) | -0.1 (0.10)

19. Primary Outcome: Change From Baseline in 10 Meter Walk or Run Velocity at Month 6: Ambulatory Participants Aged >=3 Years
Description: The 10 meter walk or run test was performed as part of NSAA. The 10 meter walk or run velocity was defined as the reciprocal of the time (in seconds) to complete the 10 meter run or walk test. The 10 meter walk or run test was performed in ambulatory children >=3 years old only as pre-specified in the protocol.
Time Frame: Baseline (Day 1) and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Meters per second
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants
Number analyzed (Participants) | 75 | 152 | 227
Meters per second | 0.2 (0.42) | -0.1 (0.27) | 0.0 (0.35)

20. Primary Outcome: Change From Baseline in 10 Meter Walk or Run Velocity at Month 12: Ambulatory Participants Aged >=3 Years
Description: as for outcome 19
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Meters per second
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants
Number analyzed (Participants) | 60 | 140 | 200
Meters per second | 0.3 (0.35) | -0.1 (0.34) | -0.0 (0.40)

21. Primary Outcome: Change From Baseline in 10 Meter Walk or Run Velocity at Month 18: Ambulatory Participants Aged >=3 Years
Description: as for outcome 19
Time Frame: Baseline (Day 1) and Month 18
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Meters per second
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants
Number analyzed (Participants) | 57 | 102 | 159
Meters per second | 0.4 (0.41) | -0.3 (0.34) | -0.0 (0.50)

22. Primary Outcome: Change From Baseline in 10 Meter Walk or Run Velocity at Month 24: Ambulatory Participants Aged >=3 Years
Description: as for outcome 19
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Meters per second
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants
Number analyzed (Participants) | 62 | 109 | 171
Meters per second | 0.5 (0.41) | -0.4 (0.39) | -0.1 (0.56)

23. Primary Outcome: Change From Baseline in 10 Meter Walk or Run Velocity at Month 30: Ambulatory Participants Aged >=3 Years
Description: as for outcome 19
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Meters per second
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants
Number analyzed (Participants) | 22 | 63 | 85
Meters per second | 0.4 (0.52) | -0.6 (0.44) | -0.3 (0.62)

24. Primary Outcome: Change From Baseline in Knee Extension of Muscle Strength at Month 6: Participants Aged >=5 Years
Description: Muscle strength was recorded by handheld myometry. Left and right knee extension was analyzed. The muscle strength test was only performed in participants >=5 years old as pre-specified in protocol.
Time Frame: Baseline (Day 1) and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 23 | 158 | 181 | 5 | 186
Kilograms
  Left Knee Extension | 0.5 (1.91) | 0.0 (1.43) | 0.1 (1.50) | 0.3 (0.29) | 0.1 (1.49)
  Right Knee Extension | 0.7 (2.35) | -0.1 (1.78) | 0.0 (1.87) | -0.0 (0.37) | 0.0 (1.85)

25. Primary Outcome: Change From Baseline in Knee Extension of Muscle Strength at Month 12: Participants Aged >=5 Years
Description: as for outcome 24
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 18 | 157 | 175 | 28 | 203
Kilograms
  Left Knee Extension | -0.1 (1.25) | -0.1 (1.85) | -0.1 (1.80) | -0.3 (1.31) | -0.1 (1.74)
  Right Knee Extension | 0.1 (1.50) | -0.4 (1.87) | -0.4 (1.84) | -0.3 (1.10) | -0.4 (1.75)

26. Primary Outcome: Change From Baseline in Knee Extension of Muscle Strength at Month 18: Participants Aged >=5 Years
Description: as for outcome 24
Time Frame: Baseline (Day 1) and Month 18
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 18 | 111 | 129 | 4 | 133
Kilograms
  Left Knee Extension | 0.7 (1.69) | -0.4 (1.95) | -0.3 (1.95) | -0.7 (1.05) | -0.3 (1.93)
  Right Knee Extension | 0.5 (1.96) | -0.7 (2.29) | -0.6 (2.28) | -0.8 (0.42) | -0.6 (2.25)

27. Primary Outcome: Change From Baseline in Knee Extension of Muscle Strength at Month 24: Participants Aged >=5 Years
Description: as for outcome 24
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 19 | 136 | 155 | 23 | 178
Kilograms
  Left Knee Extension | -0.4 (2.37) | -0.6 (1.95) | -0.6 (2.00) | -0.5 (1.64) | -0.6 (1.95)
  Right Knee Extension | 0.0 (2.77) | -1.0 (2.13) | -0.9 (2.23) | -0.7 (1.62) | -0.8 (2.16)

28. Primary Outcome: Change From Baseline in Knee Extension of Muscle Strength at Month 30: Participants Aged >=5 Years
Description: as for outcome 24
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 7 | 76 | 83 | 3 | 86
Kilograms
  Left Knee Extension | -0.9 (2.12) | -0.7 (2.66) | -0.7 (2.60) | -0.4 (0.36) | -0.7 (2.56)
  Right Knee Extension | -2.3 (2.89) | -1.4 (2.76) | -1.4 (2.76) | -1.1 (0.44) | -1.4 (2.72)

29. Primary Outcome: Change From Baseline in Elbow Flexion of Muscle Strength at Month 6: Participants Aged >=5 Years
Description: Muscle strength was recorded by handheld myometry. Left and right elbow flexion were analyzed. The muscle strength test was only performed in participants >=5 years old as pre-specified in the protocol.
Time Frame: Baseline (Day 1) and Month 6
Population: Full Analysis Set included all participants who had been enrolled in the study. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure. 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 24 | 160 | 184 | 5 | 189
Kilograms
  Left Elbow Flexion | 0.3 (0.85) | 0.3 (0.93) | 0.3 (0.92) | -0.4 (0.30) | 0.3 (0.92)
  Right Elbow Flexion: number analyzed (Participants) | 24 | 159 | 183 | 5 | 188
  Right Elbow Flexion | 0.4 (0.81) | 0.3 (0.93) | 0.3 (0.91) | -0.3 (0.25) | 0.3 (0.91)

30. Primary Outcome: Change From Baseline in Elbow Flexion of Muscle Strength at Month 12: Participants Aged >=5 Years
Description: as for outcome 29
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 19 | 159 | 178 | 29 | 207
Kilograms
  Left Elbow Flexion | 0.5 (0.97) | 0.1 (1.02) | 0.2 (1.02) | 0.1 (1.12) | 0.1 (1.03)
  Right Elbow Flexion: number analyzed (Participants) | 19 | 158 | 177 | 29 | 206
  Right Elbow Flexion | 0.5 (0.79) | 0.2 (1.07) | 0.3 (1.05) | -0.1 (0.89) | 0.2 (1.03)

31. Primary Outcome: Change From Baseline in Elbow Flexion of Muscle Strength at Month 18: Participants Aged >=5 Years
Description: as for outcome 29
Time Frame: Baseline (Day 1) and Month 18
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 19 | 114 | 133 | 4 | 137
Kilograms
  Left Elbow Flexion | 0.7 (0.80) | 0.2 (1.14) | 0.2 (1.11) | -1.0 (0.83) | 0.2 (1.12)
  Right Elbow Flexion: number analyzed (Participants) | 19 | 113 | 132 | 3 | 135
  Right Elbow Flexion | 0.5 (0.85) | 0.2 (1.16) | 0.3 (1.12) | -0.9 (1.35) | 0.2 (1.13)

32. Primary Outcome: Change From Baseline in Elbow Flexion of Muscle Strength at Month 24: Participants Aged >=5 Years
Description: as for outcome 29
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 20 | 137 | 157 | 23 | 180
Kilograms
  Left Elbow Flexion | 0.8 (0.89) | 0.0 (1.18) | 0.1 (1.17) | -0.0 (0.92) | 0.1 (1.14)
  Right Elbow Flexion | 0.9 (0.81) | 0.1 (1.16) | 0.2 (1.15) | -0.3 (1.15) | 0.1 (1.16)

33. Primary Outcome: Change From Baseline in Elbow Flexion of Muscle Strength at Month 30: Participants Aged >=5 Years
Description: as for outcome 29
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 7 | 77 | 84 | 4 | 88
Kilograms
  Left Elbow Flexion | 0.8 (0.72) | 0.2 (1.58) | 0.2 (1.53) | -0.0 (0.83) | 0.2 (1.51)
  Right Elbow Flexion | 0.4 (0.70) | 0.4 (1.56) | 0.4 (1.50) | -0.0 (0.68) | 0.4 (1.47)

34. Primary Outcome: Change From Baseline in Elbow Extension of Muscle Strength at Month 6: Participants Aged >=5 Years
Description: Muscle strength was recorded by handheld myometry. Left and right elbow extension were analyzed. The muscle strength test was only performed in participants >=5 years old as pre-specified in protocol.
Time Frame: Baseline (Day 1) and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 23 | 160 | 183 | 5 | 188
Kilograms
  Left Elbow Extension | 0.4 (0.85) | 0.2 (0.78) | 0.2 (0.79) | 0.1 (0.21) | 0.2 (0.78)
  Right Elbow Extension | 0.3 (1.22) | 0.3 (0.87) | 0.3 (0.92) | 0.1 (0.26) | 0.3 (0.91)

35. Primary Outcome: Change From Baseline in Elbow Extension Muscle Strength at Month 12: Participants Aged >=5 Years
Description: as for outcome 34
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 18 | 159 | 177 | 29 | 206
Kilograms
  Left Elbow Extension | 0.2 (0.74) | 0.2 (0.87) | 0.2 (0.85) | 0.0 (0.68) | 0.2 (0.83)
  Right Elbow Extension | 0.4 (0.88) | 0.3 (0.97) | 0.3 (0.96) | 0.2 (0.76) | 0.3 (0.93)

36. Primary Outcome: Change From Baseline in Elbow Extension Muscle Strength at Month 18: Participants Aged >=5 Years
Description: as for outcome 34
Time Frame: Baseline (Day 1) and Month 18
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 18 | 114 | 132 | 4 | 136
Kilograms
  Left Elbow Extension | 0.6 (0.80) | 0.2 (1.00) | 0.2 (0.99) | -0.4 (0.73) | 0.2 (0.98)
  Right Elbow Extension | -0.0 (0.84) | 0.2 (1.09) | 0.2 (1.06) | -0.2 (0.13) | 0.2 (1.04)

37. Primary Outcome: Change From Baseline in Elbow Extension Muscle Strength at Month 24: Participants Aged >=5 Years
Description: as for outcome 34
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 19 | 137 | 156 | 23 | 179
Kilograms
  Left Elbow Extension | 1.1 (1.14) | 0.1 (1.03) | 0.3 (1.08) | -0.1 (0.73) | 0.2 (1.05)
  Right Elbow Extension | 0.7 (1.29) | 0.0 (1.09) | 0.1 (1.13) | 0.3 (0.96) | 0.1 (1.11)

38. Primary Outcome: Change From Baseline in Elbow Extension Muscle Strength at Month 30: Participants Aged >=5 Years
Description: as for outcome 34
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Groups:
- Total Participants: Participants diagnosed with DMD who were ambulant and and who were non-ambulatory (i.e., used wheel chair full-time or were unable to complete daily activities [such as going to bathroom] by walking independently, based on performance reported at home by participant or caregiver and verification by trained CE with the inability to perform the 10-meter run/walk assessment) were included.
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 7 | 77 | 84 | 4 | 88
Kilograms
  Left Elbow Extension | 0.8 (1.55) | 0.2 (1.30) | 0.3 (1.32) | -0.3 (0.79) | 0.3 (1.30)
  Right Elbow Extension | -0.9 (0.72) | 0.3 (1.37) | 0.2 (1.36) | -0.0 (0.37) | 0.2 (1.33)

39. Primary Outcome: Change From Baseline in Shoulder Abduction of Muscle Strength at Month 6: Participants Aged >=5 Years
Description: Muscle strength was recorded by handheld myometry. Left and right shoulder abduction were analyzed. The muscle strength test was only performed in participants >=5 years old as pre-specified in the protocol.
Time Frame: Baseline (Day 1) and Month 6
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 24 | 159 | 183 | 5 | 188
Kilograms
  Left Shoulder Abduction: number analyzed (Participants) | 23 | 159 | 182 | 5 | 187
  Left Shoulder Abduction | 0.4 (1.15) | 0.4 (0.87) | 0.4 (0.91) | -0.1 (0.45) | 0.4 (0.90)
  Right Shoulder Abduction | 0.5 (0.95) | 0.4 (0.90) | 0.4 (0.90) | 0.3 (0.10) | 0.4 (0.89)

40. Primary Outcome: Change From Baseline in Shoulder Abduction of Muscle Strength at Month 12: Participants Aged >=5 Years
Description: as for outcome 39
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 19 | 158 | 177 | 29 | 206
Kilograms
  Left Shoulder Abduction: number analyzed (Participants) | 18 | 158 | 176 | 29 | 205
  Left Shoulder Abduction | 0.5 (0.76) | 0.4 (0.89) | 0.4 (0.88) | 0.1 (0.82) | 0.4 (0.88)
  Right Shoulder Abduction | 0.6 (0.86) | 0.5 (1.00) | 0.5 (0.99) | 0.1 (0.97) | 0.4 (0.99)

41. Primary Outcome: Change From Baseline in Shoulder Abduction of Muscle Strength at Month 18: Participants Aged >=5 Years
Description: as for outcome 39
Time Frame: Baseline (Day 1) and Month 18
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 19 | 113 | 132 | 4 | 136
Kilograms
  Left Shoulder Abduction: number analyzed (Participants) | 18 | 113 | 131 | 4 | 135
  Left Shoulder Abduction | 0.5 (0.65) | 0.4 (0.98) | 0.4 (0.94) | -1.0 (0.60) | 0.3 (0.96)
  Right Shoulder Abduction | 0.8 (0.98) | 0.4 (1.05) | 0.5 (1.04) | -0.8 (0.55) | 0.4 (1.05)

42. Primary Outcome: Change From Baseline in Shoulder Abduction of Muscle Strength at Month 24: Participants Aged >=5 Years
Description: as for outcome 39
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 20 | 136 | 156 | 23 | 179
Kilograms
  Left Shoulder Abduction: number analyzed (Participants) | 19 | 136 | 155 | 23 | 178
  Left Shoulder Abduction | 1.1 (1.04) | 0.3 (1.13) | 0.4 (1.15) | 0.0 (0.80) | 0.4 (1.12)
  Right Shoulder Abduction | 1.2 (1.11) | 0.6 (1.25) | 0.6 (1.24) | -0.1 (1.04) | 0.5 (1.24)

43. Primary Outcome: Change From Baseline in Shoulder Abduction of Muscle Strength at Month 30: Participants Aged >=5 Years
Description: as for outcome 39
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 7 | 76 | 83 | 4 | 87
Kilograms
  Left Shoulder Abduction | 0.6 (1.28) | 0.6 (1.25) | 0.6 (1.25) | 0.8 (1.00) | 0.6 (1.23)
  Right Shoulder Abduction | 0.8 (0.93) | 0.8 (1.34) | 0.8 (1.31) | 1.3 (1.77) | 0.8 (1.32)

44. Primary Outcome: Change From Baseline in Range of Motion (ROM) at Bilateral Ankles at Month 6
Description: Range of motion was evaluated by using goniometry to record any occurrences of ankle contractures. The ROM at left and right ankles were measured in degrees of passive dorsiflexion.
Time Frame: Baseline (Day 1) and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Degrees of passive dorsiflexion
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 94 | 162 | 256 | 5 | 261
Degrees of passive dorsiflexion
  Left Ankle Joint | -0.5 (9.12) | 0.8 (10.94) | 0.3 (10.31) | -8.2 (8.50) | 0.2 (10.33)
  Right Ankle Joint | -1.2 (8.59) | -0.4 (10.69) | -0.7 (9.96) | -8.2 (5.45) | -0.8 (9.94)

45. Primary Outcome: Change From Baseline in ROM at Bilateral Ankles at Month 12
Description: as for outcome 44
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Degrees of passive dorsiflexion
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 80 | 160 | 240 | 28 | 268
Degrees of passive dorsiflexion
  Left Ankle Joint | -2.6 (10.13) | -2.0 (11.06) | -2.2 (10.74) | -11.6 (18.18) | -3.2 (12.05)
  Right Ankle Joint | -3.1 (9.19) | -2.8 (10.85) | -2.9 (10.31) | -7.9 (19.74) | -3.4 (11.70)

46. Primary Outcome: Change From Baseline in ROM at Bilateral Ankles at Month 18
Description: as for outcome 44
Time Frame: Baseline (Day 1) and Month 18
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Degrees of passive dorsiflexion
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 77 | 115 | 192 | 4 | 196
Degrees of passive dorsiflexion
  Left Ankle Joint | -1.8 (9.19) | -4.0 (10.90) | -3.1 (10.28) | -8.8 (12.47) | -3.2 (10.32)
  Right Ankle Joint | -2.2 (8.91) | -4.5 (11.50) | -3.6 (10.58) | -5.0 (4.24) | -3.6 (10.48)

47. Primary Outcome: Change From Baseline in ROM at Bilateral Ankles at Month 24
Description: as for outcome 44
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Degrees of passive dorsiflexion
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 75 | 136 | 211 | 23 | 234
Degrees of passive dorsiflexion
  Left Ankle Joint | -2.8 (8.59) | -4.8 (12.09) | -4.1 (11.00) | -8.5 (15.79) | -4.6 (11.59)
  Right Ankle Joint | -3.6 (8.78) | -6.0 (12.88) | -5.1 (11.62) | -11.4 (15.77) | -5.8 (12.20)

48. Primary Outcome: Change From Baseline in ROM at Bilateral Ankles at Month 30
Description: as for outcome 44
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Degrees of passive dorsiflexion
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 30 | 76 | 106 | 4 | 110
Degrees of passive dorsiflexion
  Left Ankle Joint | 0.3 (9.50) | -4.9 (12.23) | -3.4 (11.71) | -4.8 (14.08) | -3.5 (11.73)
  Right Ankle Joint | 0.1 (8.08) | -6.5 (13.04) | -4.6 (12.18) | -2.5 (6.24) | -4.5 (12.01)

49. Primary Outcome: Change From Baseline in ROM at Bilateral Elbows at Month 6
Description: Range of motion was evaluated by using goniometry to record any occurrences of elbow contractures. The ROM at left and right elbows were measured in degrees of passive extension.
Time Frame: Baseline (Day 1) and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Degrees of passive extension
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 94 | 162 | 256 | 5 | 261
Degrees of passive extension
  Right Elbow Joint | 1.0 (7.13) | 1.0 (6.82) | 1.0 (6.92) | -3.2 (7.79) | 0.9 (6.95)
  Left Elbow Joint | 0.8 (7.13) | 0.7 (6.17) | 0.8 (6.53) | -4.0 (2.92) | 0.7 (6.51)

50. Primary Outcome: Change From Baseline in ROM at Bilateral Elbows at Month 12
Description: as for outcome 49
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Degrees of passive extension
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 80 | 160 | 240 | 29 | 269
Degrees of passive extension
  Right Elbow Joint | -2.7 (9.86) | -0.3 (7.85) | -1.1 (8.63) | -2.7 (11.19) | -1.3 (8.93)
  Left Elbow Joint | -2.3 (10.33) | -1.3 (7.90) | -1.6 (8.77) | -3.3 (11.52) | -1.8 (9.10)

51. Primary Outcome: Change From Baseline in ROM at Bilateral Elbows at Month 18
Description: as for outcome 49
Time Frame: Baseline (Day 1) and Month 18
Population: Full Analysis Set included all participants who had been enrolled in the study. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Number Analyzed signifies participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Degrees of passive extension
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 77 | 115 | 192 | 4 | 196
Degrees of passive extension
  Right Elbow Joint: number analyzed (Participants) | 76 | 115 | 191 | 4 | 195
  Right Elbow Joint | -1.6 (8.44) | -1.8 (8.03) | -1.7 (8.18) | -7.0 (12.99) | -1.8 (8.28)
  Left Elbow Joint | -1.1 (8.43) | -2.6 (6.41) | -2.0 (7.30) | -10.3 (2.63) | -2.1 (7.33)

52. Primary Outcome: Change From Baseline in ROM at Bilateral Elbows at Month 24
Description: as for outcome 49
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Degrees of passive extension
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 75 | 137 | 212 | 23 | 235
Degrees of passive extension
  Right Elbow Joint | 0.1 (6.68) | -1.0 (7.42) | -0.6 (7.17) | -5.1 (13.22) | -1.1 (8.04)
  Left Elbow Joint | 0.7 (6.79) | -1.5 (6.99) | -0.7 (6.98) | -5.7 (13.87) | -1.2 (8.02)

53. Primary Outcome: Change From Baseline in ROM at Bilateral Elbows at Month 30
Description: as for outcome 49
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Degrees of passive extension
Groups:
- Total Participants: Participants diagnosed with DMD who were ambulant and time of screening and who were non-ambulatory (i.e., used wheel chair full-time or were unable to complete daily activities [such as going to bathroom] by walking independently, based on performance reported at home by participant or caregiver and verification by trained CE with the inability to perform the 10-meter run/walk assessment) were included.
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 30 | 77 | 107 | 4 | 111
Degrees of passive extension
  Right Elbow Joint | 1.0 (5.47) | -1.9 (7.52) | -1.1 (7.10) | -5.0 (17.74) | -1.2 (7.60)
  Left Elbow Joint | 1.0 (6.69) | -2.2 (7.23) | -1.3 (7.19) | -9.0 (14.26) | -1.5 (7.58)

54. Primary Outcome: Change From Baseline in Percent Predicted Forced Vital Capacity (%pFVC) at Month 12: Participants Aged >=6 Years
Description: Forced vital capacity (FVC) is the volume of air that can be maximally forcefully exhaled after taking the deepest breath possible and was measured using spirometry. The percent predicted FVC was calculated from FVC (measured in liter) according to age, height (estimated height as derived from the ulna length for non-ambulatory participants), ethnicity, and gender using multi-ethnic reference values for spirometry. The pulmonary function assessments were performed in participants aged >=6 years as pre-specified in the protocol.
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent predicted FVC
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 158 | 30 | 188
Percent predicted FVC | -2.9 (15.85) | -5.7 (19.79) | -3.4 (16.52)

55. Primary Outcome: Change From Baseline in %pFVC at Month 24: Participants Aged >=6 Years
Description: FVC is the volume of air that can be maximally forcefully exhaled after taking the deepest breath possible and was measured using spirometry. The percent predicted FVC was calculated from FVC (measured in liter) according to age, height (estimated height as derived from the ulna length for non-ambulatory participants), ethnicity, and gender using multi-ethnic reference values for spirometry. The pulmonary function assessments were performed in participants aged >=6 years as pre-specified in the protocol.
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent predicted FVC
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 135 | 23 | 158
Percent predicted FVC | -4.3 (15.97) | -14.1 (20.68) | -5.7 (17.02)

56. Primary Outcome: Change From Baseline in %pFVC at Month 30: Participants Aged >=6 Years
Description: as for outcome 55
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent predicted FVC
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 75 | 4 | 79
Percent predicted FVC | 105.4 (975.57) | -3.2 (9.41) | 99.9 (950.53)

57. Primary Outcome: Change From Baseline in %pFVC at Month 12: Participants Aged >=6 Years (Unplanned Analysis)
Description: FVC is the volume of air that can be maximally forcefully exhaled after taking the deepest breath possible and was measured using spirometry. The percent predicted FVC was calculated from FVC (measured in liter) according to age, height (estimated height as derived from the ulna length for non-ambulatory participants), ethnicity, and gender using multi-ethnic reference values for spirometry. The pulmonary function assessments were performed in participants aged >=6 years as pre-specified in the protocol. Incorrect data were addressed by unplanned analysis.
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent predicted FVC
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 158 | 30 | 188
Percent predicted FVC | -2.9 (15.85) | -5.7 (19.79) | -3.4 (16.52)

58. Primary Outcome: Change From Baseline in %pFVC at Month 24: Participants Aged >=6 Years (Unplanned Analysis)
Description: as for outcome 57
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent predicted FVC
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 135 | 23 | 158
Percent predicted FVC | -4.3 (15.97) | -14.1 (20.68) | -5.7 (17.02)

59. Primary Outcome: Change From Baseline in %pFVC at Month 30: Participants Aged >=6 Years (Unplanned Analysis)
Description: as for outcome 57
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent predicted FVC
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 74 | 4 | 78
Percent predicted FVC | -7.2 (16.41) | -3.2 (9.41) | -7.0 (16.12)

60. Primary Outcome: Change From Baseline in Percent Predicted Forced Expiratory Volume in One Second (%pFEV1) at Month 12: Participants Aged >=6 Years
Description: Forced expiratory volume in one second (FEV1) is the volume of air forcefully exhaled in 1 second and was measured using spirometry. The %pFEV1 was calculated from FEV1 (measured in liter) according to age, height (estimated height as derived from the ulna length for non-ambulatory participants), ethnicity, and gender using multi-ethnic reference values for Spirometry. The pulmonary function assessments were performed only in participants >=6 years old as pre-specified in protocol.
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent predicted FEV1
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 158 | 30 | 188
Percent predicted FEV1 | -1.8 (18.65) | -4.0 (19.64) | -2.1 (18.78)

61. Primary Outcome: Change From Baseline in %pFEV1 at Month 24: Participants Aged >=6 Years
Description: FEV1 is the volume of air forcefully exhaled in 1 second and was measured using spirometry. The %pFEV1 was calculated from FEV1 (measured in liter) according to age, height (estimated height as derived from the ulna length for non-ambulatory participants), ethnicity, and gender using multi-ethnic reference values for Spirometry. The pulmonary function assessments were performed only in participants >=6 years old as pre-specified in protocol.
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent predicted FEV1
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 135 | 23 | 158
Percent predicted FEV1 | -3.9 (19.38) | -10.2 (20.94) | -4.8 (19.67)

62. Primary Outcome: Change From Baseline in %pFEV1 at Month 30: Participants Aged >=6 Years
Description: as for outcome 61
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent predicted FEV1
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 75 | 4 | 79
Percent predicted FEV1 | 115.2 (1037.35) | -5.8 (8.83) | 109.1 (1010.75)

63. Primary Outcome: Change From Baseline in %pFEV1 at Month 12: Participants Aged >=6 Years (Unplanned Analysis)
Description: FEV1 is the volume of air forcefully exhaled in 1 second and was measured using spirometry. The %pFEV1 was calculated from FEV1 (measured in liter) according to age, height (estimated height as derived from the ulna length for non-ambulatory participants), ethnicity, and gender using multi-ethnic reference values for Spirometry. The pulmonary function assessments were performed only in participants >=6 years old as pre-specified in protocol. Incorrect data were addressed by unplanned analysis.
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent predicted FEV1
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 158 | 30 | 188
Percent predicted FEV1 | -1.8 (18.65) | -4.0 (19.64) | -2.1 (18.78)

64. Primary Outcome: Change From Baseline in %pFEV1 at Month 24: Participants Aged >=6 Years (Unplanned Analysis)
Description: as for outcome 63
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent predicted FEV1
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 135 | 23 | 158
Percent predicted FEV1 | -3.9 (19.38) | -10.2 (20.94) | -4.8 (19.67)

65. Primary Outcome: Change From Baseline in %pFEV1 at Month 30: Participants Aged >=6 Years (Unplanned Analysis)
Description: as for outcome 63
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent predicted FEV1
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 74 | 4 | 78
Percent predicted FEV1 | -4.6 (18.97) | -5.8 (8.83) | -4.6 (18.56)

66. Primary Outcome: Change From Baseline in Maximum Inspiratory Pressure at Month 12: Participants Aged >=6 Years
Description: The pulmonary function assessments were performed only in participants >=6 years old as pre-specified in protocol.
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Centimeter of water (cm H2O)
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 141 | 28 | 169
Centimeter of water (cm H2O) | 1.4 (18.22) | -3.1 (20.46) | 0.6 (18.62)

67. Primary Outcome: Change From Baseline in Maximum Inspiratory Pressure at Month 24: Participants Aged >=6 Years
Description: The pulmonary function assessments were performed only in participants >=6 years old as pre-specified in protocol.
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Centimeter of water (cm H2O)
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 122 | 23 | 145
Centimeter of water (cm H2O) | 0.9 (18.24) | -2.8 (17.24) | 0.3 (18.08)

68. Primary Outcome: Change From Baseline in Maximum Inspiratory Pressure at Month 30: Participants Aged >=6 Years
Description: The pulmonary function assessments were performed only in participants >=6 years old as pre-specified in protocol.
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Centimeter of water (cm H2O)
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 67 | 4 | 71
Centimeter of water (cm H2O) | 2.5 (19.19) | -14.0 (13.22) | 1.6 (19.22)

69. Primary Outcome: Change From Baseline in Maximum Expiratory Pressure at Month 12: Participants Aged >=6 Years
Description: The pulmonary function assessments were performed only in participants >=6 years old as pre-specified in SAP.
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Centimeter of water (cm H2O)
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 154 | 29 | 183
Centimeter of water (cm H2O) | 1.0 (14.72) | -5.5 (14.24) | -0.0 (14.80)

70. Primary Outcome: Change From Baseline in Maximum Expiratory Pressure at Month 24: Participants Aged >=6 Years
Description: The pulmonary function assessments were performed only in participants >=6 years old as pre-specified in SAP.
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Centimeter of water (cm H2O)
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 132 | 23 | 155
Centimeter of water (cm H2O) | 0.6 (18.07) | -2.5 (13.67) | 0.1 (17.48)

71. Primary Outcome: Change From Baseline in Maximum Expiratory Pressure at Month 30: Participants Aged >=6 Years
Description: The pulmonary function assessments were performed only in participants >=6 years old as pre-specified in SAP.
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Centimeter of water (cm H2O)
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 75 | 4 | 79
Centimeter of water (cm H2O) | 1.7 (17.91) | -20.3 (23.61) | 0.6 (18.68)

72. Primary Outcome: Change From Baseline in Peak Cough Flow at Month 12: Participants Aged >=6 Years
Description: The pulmonary function assessments were performed only in participants >=6 years old as pre-specified in protocol.
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters per minute
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 157 | 30 | 187
Liters per minute | 14.0 (46.61) | 38.6 (61.50) | 17.9 (49.94)

73. Primary Outcome: Change From Baseline in Peak Cough Flow at Month 24: Participants Aged >=6 Years
Description: The pulmonary function assessments were performed only in participants >=6 years old as pre-specified in protocol.
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters per minute
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 133 | 23 | 156
Liters per minute | 20.7 (59.04) | 46.1 (67.78) | 24.4 (60.84)

74. Primary Outcome: Change From Baseline in Peak Cough Flow at Month 30: Participants Aged >=6 Years
Description: The pulmonary function assessments were performed only in participants >=6 years old as pre-specified in protocol.
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters per minute
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 74 | 4 | 78
Liters per minute | 25.2 (62.83) | 74.0 (24.84) | 27.7 (62.32)

75. Primary Outcome: Change From Baseline in Peak Cough Flow at Month 12: Participants Aged >=6 Years (Unplanned Analysis)
Description: The pulmonary function assessments were performed only in participants >=6 years old as pre-specified in protocol. Incorrect data were addressed by unplanned analysis.
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters per minute
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 157 | 30 | 187
Liters per minute | 14.0 (46.61) | 38.6 (61.50) | 17.9 (49.94)

76. Primary Outcome: Change From Baseline in Peak Cough Flow at Month 24: Participants Aged >=6 Years (Unplanned Analysis)
Description: as for outcome 75
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters per minute
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 132 | 23 | 155
Liters per minute | 22.4 (55.94) | 46.1 (67.78) | 25.9 (58.22)

77. Primary Outcome: Change From Baseline in Peak Cough Flow at Month 30: Participants Aged >=6 Years (Unplanned Analysis)
Description: as for outcome 75
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters per minute
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 74 | 4 | 78
Liters per minute | 25.2 (62.83) | 74.0 (24.84) | 27.7 (62.32)

78. Primary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) at Month 12: Participants Aged >=6 Years
Description: LVEF was the percentage of blood that was ejected out of left ventricle with each contraction, estimated by echocardiography. The LVEF was only performed in participants >=6 years old as pre-specified in protocol.
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of ejected blood
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 160 | 29 | 189
Percentage of ejected blood | 4.1 (45.37) | -0.4 (6.32) | 3.4 (41.83)

79. Primary Outcome: Change From Baseline in LVEF at Month 24: Participants Aged >=6 Years
Description: as for outcome 78
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of ejected blood
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 137 | 24 | 161
Percentage of ejected blood | -0.7 (5.43) | -1.6 (7.58) | -0.8 (5.78)

80. Primary Outcome: Change From Baseline in LVEF at Month 30: Participants Aged >=6 Years
Description: as for outcome 78
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of ejected blood
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 78 | 4 | 82
Percentage of ejected blood | -0.3 (6.42) | -2.0 (4.69) | -0.4 (6.34)

81. Primary Outcome: Change From Baseline in LVEF at Month 12: Participants Aged >=6 Years (Unplanned Analysis)
Description: LVEF was the percentage of blood that was ejected out of left ventricle with each contraction, estimated by echocardiography. The LVEF was only performed in participants >=6 years old as pre-specified in protocol. Incorrect data were addressed by unplanned analysis.
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of ejected blood
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 159 | 29 | 188
Percentage of ejected blood | 0.5 (6.27) | -0.4 (6.32) | 0.4 (6.27)

82. Primary Outcome: Change From Baseline in LVEF at Month 24: Participants Aged >=6 Years (Unplanned Analysis)
Description: as for outcome 81
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of ejected blood
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 137 | 24 | 161
Percentage of ejected blood | -0.7 (5.43) | -1.6 (7.58) | -0.8 (5.78)

83. Primary Outcome: Change From Baseline in LVEF at Month 30: Participants Aged >=6 Years (Unplanned Analysis)
Description: as for outcome 81
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of ejected blood
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 78 | 4 | 82
Percentage of ejected blood | -0.3 (6.42) | -2.0 (4.69) | -0.4 (6.34)

84. Primary Outcome: Change From Baseline in Wechsler Intelligence Scale for Children (WISC)-IV Score at Month 24: Ambulatory Participants >= 6 to <=16 Years
Description: WISC-IV is an individually administered intelligence test for children between the ages of 6 and 16. The WISC-IV Composites are: Verbal Comprehension, Perceptual Reasoning, Working Memory, and Processing Speed. Scores from the Composites constitute the WISC-IV Full Scale IQ score which ranges from 40 (Exceptionally Low) to 160 (Exceptionally Superior), higher scores indicated more intelligence. The WISC was only performed in ambulatory participants >= 6 to <=16 years old as pre-specified in the protocol.
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age >=6 Years
Number analyzed (Participants) | 97
Units on a scale | 1.0 (8.59)

85. Secondary Outcome: Number of Participants With Type of DMD Mutation
Description: Number of participants as per type of mutation: exon deletion, exon duplication, point mutation, small insertion, small deletion and others is presented in this outcome measure. One participant could have more than 1 mutation type.
Time Frame: Up to Month 30
Population: Full Analysis Set included all participants who had been enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 177 | 36 | 312
Participants
  Exon Deletion | 64 | 127 | 18 | 209
  Exon Duplication | 10 | 21 | 6 | 37
  Point Mutation | 18 | 21 | 8 | 47
  Small Insertion | 1 | 1 | 3 | 5
  Small Deletion | 5 | 7 | 1 | 13
  Others | 2 | 1 | 0 | 3

86. Secondary Outcome: Number of Participants With Each Affected Exon by Mutation Types
Description: Number of participants with each affected exon by mutation types is presented in this outcome measure. Only those categories with non-zero values have been reported.
Time Frame: Up to Month 30
Population: Full Analysis Set included all participants who had been enrolled in the study. 'Number of Participants Analyzed' signifies all participants in the Full Analysis Set with affected exon. The frequency (count) of each affected exon by mutation types was defined to be plotted for 3 groups combined, because the mutation types/affected exons were not anticipated to be varied in different age groups or by ambulation status according to available evidence globally.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Participants
Number analyzed (Participants) | 299
Participants
  Exon 1, Exon deletion | 3
  Exon 2, Exon deletion | 3
  Exon 2, Exon duplication | 6
  Exon 3, Exon deletion | 16
  Exon 3, Exon duplication | 5
  Exon 4, Exon deletion | 16
  Exon 4, Exon duplication | 5
  Exon 5, Exon deletion | 21
  Exon 5, Exon duplication | 7
  Exon 5, Point Mutation | 1
  Exon 6, Exon deletion | 20
  Exon 6, Exon duplication | 8
  Exon 6, Point Mutation | 1
  Exon 6, Others | 1
  Exon 7, Exon deletion | 20
  Exon 7, Exon duplication | 8
  Exon 8, Exon deletion | 21
  Exon 8, Exon duplication | 6
  Exon 9, Exon deletion | 21
  Exon 9, Exon duplication | 5
  Exon 10, Exon deletion | 17
  Exon 10, Exon duplication | 4
  Exon 10, Point Mutation | 1
  Exon 11, Exon deletion | 17
  Exon 11, Exon duplication | 5
  Exon 12, Exon deletion | 16
  Exon 12, Exon duplication | 4
  Exon 13, Exon deletion | 17
  Exon 13, Exon duplication | 3
  Exon 13, Small deletion | 1
  Exon 14, Exon deletion | 17
  Exon 14, Exon duplication | 3
  Exon 15, Exon deletion | 17
  Exon 15, Exon duplication | 3
  Exon 15, Point Mutation | 1
  Exon 16, Exon deletion | 18
  Exon 16, Exon duplication | 3
  Exon 17, Exon deletion | 20
  Exon 17, Exon duplication | 2
  Exon 18, Exon deletion | 15
  Exon 18, Exon duplication | 3
  Exon 19, Exon deletion | 14
  Exon 19, Exon duplication | 3
  Exon 19, Point Mutation | 2
  Exon 20, Exon deletion | 13
  Exon 20, Exon duplication | 3
  Exon 20, Point Mutation | 3
  Exon 21, Exon deletion | 12
  Exon 21, Exon duplication | 3
  Exon 21, Point Mutation | 1
  Exon 22, Exon deletion | 12
  Exon 22, Exon duplication | 3
  Exon 22, Point Mutation | 1
  Exon 23, Exon deletion | 12
  Exon 23, Exon duplication | 3
  Exon 23, Point Mutation | 4
  Exon 24, Exon deletion | 12
  Exon 24, Exon duplication | 3
  Exon 24, Point Mutation | 3
  Exon 24, Small insertion | 1
  Exon 25, Exon deletion | 12
  Exon 25, Exon duplication | 3
  Exon 25, Point Mutation | 1
  Exon 25, Small deletion | 1
  Exon 26, Exon deletion | 12
  Exon 26, Exon duplication | 2
  Exon 26, Point Mutation | 3
  Exon 26, Small insertion | 1
  Exon 26, Small deletion | 1
  Exon 27, Exon deletion | 12
  Exon 27, Exon duplication | 2
  Exon 27, Point Mutation | 1
  Exon 27, Small deletion | 1
  Exon 28, Exon deletion | 12
  Exon 28, Exon duplication | 2
  Exon 28, Point Mutation | 1
  Exon 29, Exon deletion | 12
  Exon 29, Exon duplication | 2
  Exon 29, Point Mutation | 2
  Exon 30, Exon deletion | 9
  Exon 30, Exon duplication | 3
  Exon 30, Point Mutation | 2
  Exon 31, Exon deletion | 9
  Exon 31, Exon duplication | 3
  Exon 31, Point Mutation | 1
  Exon 32, Exon deletion | 9
  Exon 32, Exon duplication | 3
  Exon 32, Point Mutation | 3
  Exon 32, Small deletion | 1
  Exon 33, Exon deletion | 9
  Exon 33, Exon duplication | 3
  Exon 33, Point Mutation | 3
  Exon 33, Small deletion | 1
  Exon 34, Exon deletion | 8
  Exon 34, Exon duplication | 3
  Exon 34, Point Mutation | 1
  Exon 35, Exon deletion | 7
  Exon 35, Exon duplication | 3
  Exon 35, Point Mutation | 2
  Exon 36, Exon deletion | 7
  Exon 36, Exon duplication | 3
  Exon 36, Point Mutation | 2
  Exon 37, Exon deletion | 7
  Exon 37, Exon duplication | 4
  Exon 37, Point Mutation | 2
  Exon 38, Exon deletion | 8
  Exon 38, Exon duplication | 4
  Exon 38, Point Mutation | 1
  Exon 39, Exon deletion | 7
  Exon 39, Exon duplication | 4
  Exon 39, Point Mutation | 1
  Exon 39, Small deletion | 1
  Exon 39, Others | 1
  Exon 40, Exon deletion | 7
  Exon 40, Exon duplication | 4
  Exon 40, Point Mutation | 1
  Exon 40, Small insertion | 1
  Exon 41, Exon deletion | 7
  Exon 41, Exon duplication | 4
  Exon 41, Point Mutation | 2
  Exon 42, Exon deletion | 7
  Exon 42, Exon duplication | 3
  Exon 42, Point Mutation | 1
  Exon 43, Exon deletion | 9
  Exon 43, Exon duplication | 5
  Exon 43, Point Mutation | 1
  Exon 44, Exon deletion | 20
  Exon 44, Exon duplication | 4
  Exon 44, Point Mutation | 3
  Exon 44, Small deletion | 1
  Exon 45, Exon deletion | 42
  Exon 45, Exon duplication | 4
  Exon 46, Exon deletion | 73
  Exon 46, Exon duplication | 3
  Exon 46, Point Mutation | 1
  Exon 47, Exon deletion | 73
  Exon 47, Exon duplication | 3
  Exon 47, Point Mutation | 1
  Exon 47, Small deletion | 1
  Exon 48, Exon deletion | 83
  Exon 48, Exon duplication | 2
  Exon 48, Point Mutation | 1
  Exon 48, Small insertion | 1
  Exon 49, Exon deletion | 96
  Exon 49, Exon duplication | 2
  Exon 49, Point Mutation | 1
  Exon 50, Exon deletion | 94
  Exon 50, Exon duplication | 2
  Exon 51, Exon deletion | 64
  Exon 51, Exon duplication | 3
  Exon 52, Exon deletion | 56
  Exon 52, Exon duplication | 3
  Exon 53, Exon deletion | 24
  Exon 53, Exon duplication | 2
  Exon 53, Point Mutation | 2
  Exon 54, Exon deletion | 22
  Exon 54, Exon duplication | 4
  Exon 55, Exon deletion | 6
  Exon 55, Exon duplication | 3
  Exon 55, Point Mutation | 1
  Exon 56, Exon deletion | 2
  Exon 56, Exon duplication | 2
  Exon 56, Small deletion | 2
  Exon 57, Exon deletion | 1
  Exon 57, Exon duplication | 2
  Exon 57, Point Mutation | 2
  Exon 58, Exon duplication | 2
  Exon 58, Point Mutation | 1
  Exon 58, Small deletion | 1
  Exon 59, Exon duplication | 2
  Exon 59, Point Mutation | 1
  Exon 60, Exon duplication | 2
  Exon 61, Exon duplication | 2
  Exon 62, Exon duplication | 1
  Exon 62, Point Mutation | 2
  Exon 63, Exon deletion | 1
  Exon 63, Exon duplication | 2
  Exon 64, Exon duplication | 2
  Exon 65, Exon deletion | 1
  Exon 65, Exon duplication | 3
  Exon 66, Exon duplication | 3
  Exon 67, Exon duplication | 3
  Exon 68, Exon duplication | 3
  Exon 69, Exon duplication | 2
  Exon 70, Exon duplication | 2
  Exon 70, Point Mutation | 1
  Exon 71, Exon duplication | 2
  Exon 72, Exon duplication | 1
  Exon 73, Exon duplication | 1
  Exon 74, Exon duplication | 1

87. Secondary Outcome: Number of Participants With DMD Mutations Affecting Any Exon Between Exon 9 and Exon 13 or Deletion That Affects Both Exon 29 and Exon 30
Description: Number of participants with DMD mutations affecting any exon between exon 9 and exon 13 or deletion that affects both exon 29 and exon 30 is presented in this outcome measure.
Time Frame: Up to Month 30
Population: Full Analysis Set included all participants who had been enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 177 | 36 | 312
Participants
  Any mutation affecting any exon between exon 9 and exon 13 | 11 | 20 | 2 | 33
  Deletion affects both exon 29 and exon 30 | 2 | 6 | 1 | 9

88. Secondary Outcome: Change From Baseline in Pediatric Outcomes Data Collection Instrument (PODCI) Global Functioning Scale and Each Core Scale Score (Pediatric Parent Report) at Months 6, 12, 18, 24 and 30
Description: The PODCI is a participant-reported assessment of musculoskeletal health intended for use in children and adolescents. The pediatric version was intended for completion by parents or caregivers of children <=10 years old. It included a Global Function Scale along with core scales: Upper Extremity and Physical Function Core Scale (8 items); Transfer and Basic Mobility Core Scale (11 items); Sports and Physical Functioning Core Scale (21 items); Pain/Comfort Core Scale (3 items); Happiness Core Scale (5 items). The scores of each PODCI global functioning scale and core scales are averaged over the number of items answered (omitted no entry items). Mean of the rescaled values is multiplied by a constant so that each global functioning scale and core scales has a final range of values between 0-100. The higher scores represent less disability and better functioning.
Time Frame: Baseline (Day 1) and Months 6, 12, 18, 24 and 30
Population: Full Analysis Set included all participants who had been enrolled in the study. Here, "Number of Participants Analyzed" signifies all participants in the Full Analysis Set with age <=10 years contributed data to the table; however, may not have evaluable data for every row. 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 146 | 245 | 9 | 254
Units on a scale
  Upper Extremity, Month 6: number analyzed (Participants) | 89 | 126 | 245 | 2 | 254
  Upper Extremity, Month 6 | 1.2 (9.58) | 0.3 (7.61) | 0.7 (8.47) | 16.5 (12.02) | 0.8 (8.61)
  Upper Extremity, Month 12: number analyzed (Participants) | 75 | 116 | 191 | 4 | 195
  Upper Extremity, Month 12 | 0.7 (10.90) | -1.4 (11.05) | -0.6 (11.01) | -8.3 (17.56) | -0.7 (11.17)
  Upper Extremity, Month 18: number analyzed (Participants) | 72 | 82 | 154 | 0 | 154
  Upper Extremity, Month 18 | 2.0 (10.54) | -0.3 (9.13) | 0.8 (9.85) |  | 0.8 (9.85)
  Upper Extremity, Month 24: number analyzed (Participants) | 72 | 78 | 150 | 0 | 150
  Upper Extremity, Month 24 | -0.8 (11.41) | -4.1 (11.83) | -2.5 (11.71) |  | -2.5 (11.71)
  Upper Extremity, Month 30: number analyzed (Participants) | 27 | 33 | 60 | 0 | 60
  Upper Extremity, Month 30 | 4.1 (9.90) | -2.2 (10.91) | 0.6 (10.85) |  | 0.6 (10.85)
  Transfer and Mobility, Month 6: number analyzed (Participants) | 89 | 126 | 245 | 2 | 254
  Transfer and Mobility, Month 6 | 1.5 (7.91) | -1.2 (8.59) | -0.1 (8.40) | 7.5 (14.85) | 0.0 (8.46)
  Transfer and Mobility, Month 12: number analyzed (Participants) | 75 | 116 | 191 | 4 | 195
  Transfer and Mobility, Month 12 | 1.9 (7.67) | -5.5 (14.75) | -2.6 (12.95) | -2.8 (17.02) | -2.6 (12.99)
  Transfer and Mobility, Month 18: number analyzed (Participants) | 72 | 82 | 154 | 0 | 154
  Transfer and Mobility, Month 18 | 1.6 (8.38) | -4.1 (12.12) | -1.4 (10.89) |  | -1.4 (10.89)
  Transfer and Mobility, Month 24: number analyzed (Participants) | 72 | 78 | 150 | 0 | 150
  Transfer and Mobility, Month 24 | -0.5 (8.69) | -9.8 (15.48) | -5.4 (13.47) |  | -5.4 (13.47)
  Transfer and Mobility, Month 30: number analyzed (Participants) | 27 | 33 | 60 | 0 | 60
  Transfer and Mobility, Month 30 | 1.0 (6.23) | -11.0 (17.83) | -5.6 (15.02) |  | -5.6 (15.02)
  Sports, Month 6: number analyzed (Participants) | 89 | 126 | 245 | 2 | 254
  Sports, Month 6 | 1.6 (13.79) | -1.5 (12.75) | -0.2 (13.24) | 1.0 (7.07) | -0.2 (13.19)
  Sports, Month 12: number analyzed (Participants) | 75 | 116 | 191 | 4 | 195
  Sports, Month 12 | 2.7 (14.76) | -7.5 (15.78) | -3.5 (16.14) | -4.3 (3.10) | -3.5 (15.98)
  Sports, Month 18: number analyzed (Participants) | 72 | 82 | 154 | 0 | 154
  Sports, Month 18 | 2.6 (14.05) | -7.5 (15.88) | -2.8 (15.83) |  | -2.8 (15.83)
  Sports, Month 24: number analyzed (Participants) | 72 | 78 | 150 | 0 | 150
  Sports, Month 24 | -1.1 (14.61) | -12.4 (16.74) | -7.0 (16.69) |  | -7.0 (16.69)
  Sports, Month 30: number analyzed (Participants) | 27 | 33 | 60 | 0 | 60
  Sports, Month 30 | 1.1 (10.29) | -19.9 (20.49) | -10.5 (19.64) |  | -10.5 (19.64)
  Pain, Month 6: number analyzed (Participants) | 89 | 126 | 245 | 2 | 254
  Pain, Month 6 | -0.3 (16.88) | 1.0 (19.01) | 0.5 (18.13) | 5.5 (7.78) | 0.5 (18.06)
  Pain, Month 12: number analyzed (Participants) | 75 | 116 | 191 | 4 | 195
  Pain, Month 12 | -1.4 (16.72) | -5.0 (21.95) | -3.6 (20.09) | -6.8 (14.20) | -3.7 (19.96)
  Pain, Month 18: number analyzed (Participants) | 72 | 82 | 154 | 0 | 154
  Pain, Month 18 | -2.1 (19.31) | -3.7 (20.12) | -2.9 (19.69) |  | -2.9 (19.69)
  Pain, Month 24: number analyzed (Participants) | 72 | 78 | 150 | 0 | 150
  Pain, Month 24 | -7.1 (18.46) | -8.5 (21.36) | -7.8 (19.97) |  | -7.8 (19.97)
  Pain, Month 30: number analyzed (Participants) | 27 | 33 | 60 | 0 | 60
  Pain, Month 30 | -6.4 (13.80) | -15.2 (19.27) | -11.2 (17.45) |  | -11.2 (17.45)
  Happiness, Month 6: number analyzed (Participants) | 88 | 126 | 214 | 2 | 216
  Happiness, Month 6 | 0.2 (15.69) | 0.0 (20.09) | 0.1 (18.37) | -10.0 (7.07) | -0.0 (18.32)
  Happiness, Month 12: number analyzed (Participants) | 75 | 116 | 191 | 4 | 195
  Happiness, Month 12 | 2.4 (14.41) | -5.6 (23.49) | -2.4 (20.74) | -17.5 (11.90) | -2.7 (20.69)
  Happiness, Month 18: number analyzed (Participants) | 72 | 82 | 154 | 0 | 154
  Happiness, Month 18 | 4.2 (14.59) | -4.2 (22.57) | -0.3 (19.65) |  | -0.3 (19.65)
  Happiness, Month 24: number analyzed (Participants) | 72 | 78 | 150 | 0 | 150
  Happiness, Month 24 | -4.4 (19.15) | -12.3 (21.44) | -8.5 (20.69) |  | -8.5 (20.69)
  Happiness, Month 30: number analyzed (Participants) | 27 | 33 | 60 | 0 | 60
  Happiness, Month 30 | 4.9 (12.73) | -12.8 (20.68) | -4.9 (19.54) |  | -4.9 (19.54)
  Global Function, Month 6: number analyzed (Participants) | 89 | 126 | 245 | 2 | 254
  Global Function, Month 6 | 1.0 (7.99) | -0.4 (8.65) | 0.2 (8.39) | 7.5 (10.61) | 0.3 (8.41)
  Global Function, Month 12: number analyzed (Participants) | 75 | 116 | 191 | 4 | 195
  Global Function, Month 12 | 1.0 (9.04) | -4.9 (12.12) | -2.6 (11.36) | -5.5 (6.40) | -2.7 (11.28)
  Global Function, Month 18: number analyzed (Participants) | 72 | 82 | 154 | 0 | 154
  Global Function, Month 18 | 1.1 (9.54) | -3.9 (10.05) | -1.6 (10.10) |  | -1.6 (10.10)
  Global Function, Month 24: number analyzed (Participants) | 72 | 78 | 150 | 0 | 150
  Global Function, Month 24 | -2.3 (10.32) | -8.7 (10.99) | -5.7 (11.11) |  | -5.7 (11.11)
  Global Function, Month 30: number analyzed (Participants) | 27 | 33 | 60 | 0 | 60
  Global Function, Month 30 | -0.1 (5.81) | -12.0 (13.73) | -6.7 (12.37) |  | -6.7 (12.37)

89. Secondary Outcome: Change From Baseline in PODCI Global Functioning Scale and Each Core Scale Score (Adolescent Parent Report) at Months 6, 12, 18, 24 and 30
Description: as for outcome 88
Time Frame: Baseline (Day 1) and Months 6, 12, 18, 24 and 30
Population: Full Analysis Set included all participants who had been enrolled in the study. Here, "Number of Participants Analyzed" signifies all participants in the Full Analysis Set with age between 11-18 years contributed data to the table; however, may not have evaluable data for every row. 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 31 | 27 | 58
Units on a scale
  Upper Extremity, Month 6: number analyzed (Participants) | 27 | 4 | 31
  Upper Extremity, Month 6 | -2.1 (8.82) | -18.8 (8.42) | -4.3 (10.32)
  Upper Extremity, Month 12: number analyzed (Participants) | 25 | 19 | 44
  Upper Extremity, Month 12 | -4.4 (9.24) | -2.4 (16.17) | -3.5 (12.57)
  Upper Extremity, Month 18: number analyzed (Participants) | 15 | 3 | 18
  Upper Extremity, Month 18 | -6.4 (8.34) | 1.3 (9.24) | -5.1 (8.72)
  Upper Extremity, Month 24: number analyzed (Participants) | 20 | 17 | 37
  Upper Extremity, Month 24 | -11.0 (13.47) | -7.5 (16.51) | -9.4 (14.83)
  Upper Extremity, Month 30: number analyzed (Participants) | 7 | 2 | 9
  Upper Extremity, Month 30 | -7.4 (10.21) | -8.0 (11.31) | -7.6 (9.71)
  Transfer and Mobility, Month 6: number analyzed (Participants) | 27 | 4 | 31
  Transfer and Mobility, Month 6 | -5.1 (13.87) | -5.8 (5.62) | -5.2 (13.03)
  Transfer and Mobility, Month 12: number analyzed (Participants) | 25 | 19 | 44
  Transfer and Mobility, Month 12 | -14.6 (17.24) | -9.2 (13.31) | -12.2 (15.73)
  Transfer and Mobility, Month 18: number analyzed (Participants) | 15 | 3 | 18
  Transfer and Mobility, Month 18 | -19.3 (15.26) | 5.7 (20.65) | -15.2 (18.27)
  Transfer and Mobility, Month 24: number analyzed (Participants) | 20 | 17 | 37
  Transfer and Mobility, Month 24 | -27.1 (21.79) | -10.3 (12.68) | -19.4 (19.84)
  Transfer and Mobility, Month 30: number analyzed (Participants) | 7 | 2 | 9
  Transfer and Mobility, Month 30 | -28.4 (25.83) | -1.5 (6.36) | -22.4 (25.42)
  Sports, Month 6: number analyzed (Participants) | 27 | 4 | 31
  Sports, Month 6 | -5.9 (14.24) | -3.0 (7.87) | -5.5 (13.52)
  Sports, Month 12: number analyzed (Participants) | 25 | 19 | 44
  Sports, Month 12 | -12.4 (15.44) | -5.4 (11.21) | -9.4 (14.07)
  Sports, Month 18: number analyzed (Participants) | 15 | 3 | 18
  Sports, Month 18 | -18.8 (17.62) | -4.7 (4.73) | -16.4 (16.96)
  Sports, Month 24: number analyzed (Participants) | 20 | 17 | 37
  Sports, Month 24 | -23.8 (17.52) | -2.6 (8.99) | -14.1 (17.69)
  Sports, Month 30: number analyzed (Participants) | 7 | 2 | 9
  Sports, Month 30 | -24.7 (17.74) | -9.5 (13.44) | -21.3 (17.42)
  Pain, Month 6: number analyzed (Participants) | 27 | 4 | 31
  Pain, Month 6 | -7.2 (14.64) | -0.5 (22.65) | -6.3 (15.57)
  Pain, Month 12: number analyzed (Participants) | 25 | 19 | 44
  Pain, Month 12 | -9.0 (20.31) | 11.3 (34.97) | -0.3 (29.07)
  Pain, Month 18: number analyzed (Participants) | 15 | 3 | 18
  Pain, Month 18 | -4.1 (20.30) | -10.3 (12.01) | -5.2 (19.03)
  Pain, Month 24: number analyzed (Participants) | 20 | 17 | 37
  Pain, Month 24 | -14.2 (20.41) | 4.9 (29.67) | -5.4 (26.52)
  Pain, Month 30: number analyzed (Participants) | 7 | 2 | 9
  Pain, Month 30 | -25.9 (22.04) | 9.0 (12.73) | -18.1 (24.92)
  Happiness, Month 6: number analyzed (Participants) | 27 | 4 | 31
  Happiness, Month 6 | -13.1 (19.57) | 7.5 (36.63) | -10.5 (22.71)
  Happiness, Month 12: number analyzed (Participants) | 25 | 19 | 44
  Happiness, Month 12 | -17.4 (19.43) | 1.6 (22.24) | -9.2 (22.54)
  Happiness, Month 18: number analyzed (Participants) | 15 | 3 | 18
  Happiness, Month 18 | -15.3 (16.31) | -10.0 (22.91) | -14.4 (16.88)
  Happiness, Month 24: number analyzed (Participants) | 20 | 17 | 37
  Happiness, Month 24 | -22.3 (20.23) | -2.1 (25.74) | -13.0 (24.79)
  Happiness, Month 30: number analyzed (Participants) | 7 | 2 | 9
  Happiness, Month 30 | -17.9 (24.30) | -17.5 (24.75) | -17.8 (22.79)
  Global Function, Month 6: number analyzed (Participants) | 27 | 4 | 31
  Global Function, Month 6 | -5.0 (8.34) | -7.3 (7.76) | -5.3 (8.18)
  Global Function, Month 12: number analyzed (Participants) | 25 | 19 | 44
  Global Function, Month 12 | -10.0 (9.34) | -1.5 (12.10) | -6.4 (11.32)
  Global Function, Month 18: number analyzed (Participants) | 15 | 3 | 18
  Global Function, Month 18 | -12.1 (8.56) | -2.0 (3.61) | -10.4 (8.77)
  Global Function, Month 24: number analyzed (Participants) | 20 | 17 | 37
  Global Function, Month 24 | -19.0 (12.31) | -3.8 (12.63) | -12.0 (14.48)
  Global Function, Month 30: number analyzed (Participants) | 7 | 2 | 9
  Global Function, Month 30 | -21.7 (16.19) | -2.5 (2.12) | -17.4 (16.40)

90. Secondary Outcome: Change From Baseline in PODCI Global Functioning Scale and Each Core Scale Score (Adolescent Self Report) at Months 6, 12, 18, 24 and 30
Description: as for outcome 88
Time Frame: Baseline (Day 1) and Months 6, 12, 18, 24 and 30
Population: as for outcome 89
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 31 | 27 | 58
Units on a scale
  Upper Extremity, Month 6: number analyzed (Participants) | 27 | 4 | 31
  Upper Extremity, Month 6 | -1.6 (8.15) | -1.0 (8.29) | -1.5 (8.03)
  Upper Extremity, Month 12: number analyzed (Participants) | 25 | 19 | 44
  Upper Extremity, Month 12 | -4.6 (10.10) | -3.3 (13.53) | -4.0 (11.58)
  Upper Extremity, Month 18: number analyzed (Participants) | 15 | 3 | 18
  Upper Extremity, Month 18 | 0.3 (7.14) | -5.7 (12.70) | -0.7 (8.13)
  Upper Extremity, Month 24: number analyzed (Participants) | 20 | 17 | 37
  Upper Extremity, Month 24 | -5.3 (10.93) | -5.5 (12.06) | -5.4 (11.30)
  Upper Extremity, Month 30: number analyzed (Participants) | 7 | 2 | 9
  Upper Extremity, Month 30 | -5.4 (7.16) | -2.0 (2.83) | -4.7 (6.46)
  Transfer and Mobility, Month 6: number analyzed (Participants) | 27 | 4 | 31
  Transfer and Mobility, Month 6 | -4.5 (10.71) | -2.0 (18.09) | -4.2 (11.53)
  Transfer and Mobility, Month 12: number analyzed (Participants) | 25 | 19 | 44
  Transfer and Mobility, Month 12 | -10.6 (18.20) | -6.3 (16.40) | -8.8 (17.38)
  Transfer and Mobility, Month 18: number analyzed (Participants) | 15 | 3 | 18
  Transfer and Mobility, Month 18 | -9.6 (11.78) | -9.7 (4.04) | -9.6 (10.78)
  Transfer and Mobility, Month 24: number analyzed (Participants) | 20 | 17 | 37
  Transfer and Mobility, Month 24 | -24.9 (19.56) | -7.9 (16.34) | -17.1 (19.86)
  Transfer and Mobility, Month 30: number analyzed (Participants) | 7 | 2 | 9
  Transfer and Mobility, Month 30 | -17.0 (19.71) | -10.0 (8.49) | -15.4 (17.61)
  Sports, Month 6: number analyzed (Participants) | 27 | 4 | 31
  Sports, Month 6 | -0.9 (14.11) | -2.8 (10.40) | -1.2 (13.56)
  Sports, Month 12: number analyzed (Participants) | 25 | 19 | 44
  Sports, Month 12 | -4.6 (19.60) | -3.2 (11.03) | -4.0 (16.30)
  Sports, Month 18: number analyzed (Participants) | 15 | 3 | 18
  Sports, Month 18 | -8.7 (14.39) | -2.7 (7.77) | -7.7 (13.52)
  Sports, Month 24: number analyzed (Participants) | 20 | 17 | 37
  Sports, Month 24 | -21.4 (19.71) | -8.2 (12.58) | -15.3 (17.87)
  Sports, Month 30: number analyzed (Participants) | 7 | 2 | 9
  Sports, Month 30 | -10.4 (13.45) | -1.5 (2.12) | -8.4 (12.32)
  Pain, Month 6: number analyzed (Participants) | 27 | 4 | 31
  Pain, Month 6 | -2.7 (17.96) | 5.5 (11.47) | -1.6 (17.34)
  Pain, Month 12: number analyzed (Participants) | 25 | 19 | 44
  Pain, Month 12 | 2.1 (26.07) | 8.3 (20.53) | 4.8 (23.77)
  Pain, Month 18: number analyzed (Participants) | 15 | 3 | 18
  Pain, Month 18 | -2.6 (17.19) | -7.7 (27.32) | -3.4 (18.30)
  Pain, Month 24: number analyzed (Participants) | 20 | 17 | 37
  Pain, Month 24 | -12.4 (24.21) | 4.0 (20.55) | -4.8 (23.78)
  Pain, Month 30: number analyzed (Participants) | 7 | 2 | 9
  Pain, Month 30 | 13.9 (23.10) | 0.0 (0.00) | 10.8 (20.92)
  Happiness, Month 6: number analyzed (Participants) | 27 | 4 | 31
  Happiness, Month 6 | -7.8 (23.14) | -8.8 (8.54) | -7.9 (21.71)
  Happiness, Month 12: number analyzed (Participants) | 25 | 19 | 44
  Happiness, Month 12 | -4.8 (23.34) | 2.6 (15.58) | -1.6 (20.48)
  Happiness, Month 18: number analyzed (Participants) | 15 | 3 | 18
  Happiness, Month 18 | -3.3 (17.29) | -8.3 (7.64) | -4.2 (16.02)
  Happiness, Month 24: number analyzed (Participants) | 20 | 17 | 37
  Happiness, Month 24 | -2.0 (31.47) | -10.6 (19.11) | -5.9 (26.53)
  Happiness, Month 30: number analyzed (Participants) | 7 | 2 | 9
  Happiness, Month 30 | -2.9 (16.29) | -2.5 (10.61) | -2.8 (14.60)
  Global Function, Month 6: number analyzed (Participants) | 27 | 4 | 31
  Global Function, Month 6 | -2.4 (6.62) | 0.3 (8.77) | -2.1 (6.82)
  Global Function, Month 12: number analyzed (Participants) | 25 | 19 | 44
  Global Function, Month 12 | -4.4 (12.66) | -0.9 (8.18) | -2.9 (10.98)
  Global Function, Month 18: number analyzed (Participants) | 15 | 3 | 18
  Global Function, Month 18 | -5.0 (7.52) | -6.3 (10.41) | -5.2 (7.72)
  Global Function, Month 24: number analyzed (Participants) | 20 | 17 | 37
  Global Function, Month 24 | -15.9 (12.85) | -4.2 (7.37) | -10.5 (12.07)
  Global Function, Month 30: number analyzed (Participants) | 7 | 2 | 9
  Global Function, Month 30 | -4.7 (12.46) | -3.5 (0.71) | -4.4 (10.81)

91. Secondary Outcome: Number of Participants According to Response to Each European Quality of Life (EuroQoL) 5 Dimension 3 Level (EQ-5D-3L) 5 Dimensions at Month 12
Description: EQ-5D-3L is a participant completed questionnaire designed to assess impact on health related quality of life. It is comprised of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension. EQ-5D-3L assessment was only performed in participants >= 16 years old as pre-specified in protocol.
Time Frame: Months 12
Population: Full Analysis Set included all participants who had been enrolled in the study. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure. 'Number Analyzed' signifies participants evaluable for specified rows. No ambulatory participants were >=16 years hence N=0 in arms "Ambulatory participants with aged >=6 years" and Total Ambulatory Participants".
Measure: Count of Participants; unit: Participants
Groups:
- Total Ambulatory Participants: Participants diagnosed with DMD who were ambulant and were greater than or equal to (>=6) years of age at the time of screening were included. No investigational drug was administered, and participants were allowed to take medications prescribed by their physicians, which constituted the SOC.
Arm/Group | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 0 | 0 | 6 | 6
Participants
  Mobility, no problems, Month 12 |  |  | 0 | 0
  Mobility, some problems, Month 12 |  |  | 3 | 3
  Mobility, extreme problems, Month 12 |  |  | 3 | 3
  Self-Care, no problems, Month 12 |  |  | 0 | 0
  Self-Care, some problems, Month 12 |  |  | 4 | 4
  Self-Care, extreme problems, Month 12 |  |  | 2 | 2
  Usual Activities, no problems, Month 12 |  |  | 1 | 1
  Usual Activities, some problems, Month 12 |  |  | 3 | 3
  Usual Activities, extreme problems, Month 12 |  |  | 2 | 2
  Pain/Discomfort, no problems, Month 12 |  |  | 5 | 5
  Pain/Discomfort, some problems, Month 12 |  |  | 1 | 1
  Pain/Discomfort, extreme problems, Month 12 |  |  | 0 | 0
  Anxiety/Depression, no problems, Month 12 |  |  | 5 | 5
  Anxiety/Depression, some problems, Month 12 |  |  | 1 | 1
  Anxiety/Depression, extreme problems, Month 12 |  |  | 0 | 0

92. Secondary Outcome: Number of Participants According to Response to Each EQ-5D-3L 5 Dimensions at Month 24
Description: as for outcome 91
Time Frame: Month 24
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 2 | 2 | 8 | 10
Participants
  Mobility, no problems, Month 24 | 1 | 1 | 0 | 1
  Mobility, some problems, Month 24 | 0 | 0 | 4 | 4
  Mobility, extreme problems, Month 24 | 1 | 1 | 4 | 5
  Self-Care, no problems, Month 24 | 0 | 0 | 0 | 0
  Self-Care, some problems, Month 24 | 1 | 1 | 3 | 4
  Self-Care, extreme problems, Month 24 | 1 | 1 | 5 | 6
  Usual Activities, no problems, Month 24 | 1 | 1 | 0 | 1
  Usual Activities, some problems, Month 24 | 0 | 0 | 5 | 5
  Usual Activities, extreme problems, Month 24 | 1 | 1 | 3 | 4
  Pain/Discomfort, no problems, Month 24 | 1 | 1 | 5 | 6
  Pain/Discomfort, some problems, Month 24 | 1 | 1 | 3 | 4
  Pain/Discomfort, extreme problems, Month 24 | 0 | 0 | 0 | 0
  Anxiety/Depression, no problems, Month 24 | 1 | 1 | 7 | 8
  Anxiety/Depression, some problems, Month 24 | 1 | 1 | 1 | 2
  Anxiety/Depression, extreme problems, Month 24 | 0 | 0 | 0 | 0

93. Secondary Outcome: Number of Participants According to Response to Each EQ-5D-3L 5 Dimensions at Month 30
Description: as for outcome 91
Time Frame: Month 30
Population: Full Analysis Set included all participants who had been enrolled in the study. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure. No participants were available for analysis at Month 30 in arms 'ambulatory participants with age >=6 years' and 'total ambulatory participants' hence, 'Number of Participants Analyzed' and 'Number Analyzed' were kept 0 for these arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 0 | 0 | 1 | 1
Participants
  Mobility, no problems, Month 30 |  |  | 0 | 0
  Mobility, some problems, Month 30 |  |  | 1 | 1
  Mobility, extreme problems, Month 30 |  |  | 0 | 0
  Self-Care, no problems, Month 30 |  |  | 0 | 0
  Self-Care, some problems, Month 30 |  |  | 0 | 0
  Self-Care, extreme problems, Month 30 |  |  | 1 | 1
  Usual Activities, no problems, Month 30 |  |  | 0 | 0
  Usual Activities, some problems, Month 30 |  |  | 0 | 0
  Usual Activities, extreme problems, Month 30 |  |  | 1 | 1
  Pain/Discomfort, no problems, Month 30 |  |  | 1 | 1
  Pain/Discomfort, some problems, Month 30 |  |  | 0 | 0
  Pain/Discomfort, extreme problems, Month 30 |  |  | 0 | 0
  Anxiety/Depression, no problems, Month 30 |  |  | 1 | 1
  Anxiety/Depression, some problems, Month 30 |  |  | 0 | 0
  Anxiety/Depression, extreme problems, Month 30 |  |  | 0 | 0

94. Secondary Outcome: Change From Baseline in EQ-5D-3L Visual Analogue Score (VAS) Assessment at Months 12, 24 and 30
Description: EQ-5D-3L is a participant completed questionnaire designed to assess impact on health related quality of life. EQ-VAS recorded the participant's self-rated health on a vertical scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state), where higher scores indicated better quality of life. EQ-VAS assessment was only performed in the participants >= 16 years old.
Time Frame: Baseline (Day 1) and Months 12, 24 and 30
Population: Full Analysis Set included all participants who had been enrolled in the study. Number of Participants Analyzed' signifies all participants in the Full Analysis Set with age >=16 years. 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Total Participants: Participants diagnosed with DMD who were non-ambulatory (i.e., used wheel chair full-time or were unable to complete daily activities [such as going to bathroom] by walking independently, based on performance reported at home by participant or caregiver and verification by trained CE with the inability to perform the 10-meter run/walk assessment) were included
Arm/Group | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 4 | 4
Units on a scale
  Month 12: number analyzed (Participants) | 3 | 3
  Month 12 | -4.0 (9.54) | -4.0 (9.54)
  Month 24: number analyzed (Participants) | 3 | 3
  Month 24 | -11.3 (7.37) | -11.3 (7.37)
  Month 30: number analyzed (Participants) | 1 | 1
  Month 30 | -14.0 (NA) — Standard deviation could not be calculated for single participant. | -14.0 (NA) — Standard deviation could not be calculated for single participant.

95. Secondary Outcome: Change From Baseline in EQ-5D-3L Index Score at Months 12, 24 and 30
Description: EQ-5D-3L index score, participants rated their current health state on 5 single-item dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression with each dimension having three levels of severity: 1=no problems, 2=some problems and 3=extreme problems. Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score was transformed and results in a total index score range of 0 to 1.00. Higher scores indicating a better quality of life. EQ-5D-3L was only performed in participants >= 16 years old.
Time Frame: Baseline (Day 1) and Months 12, 24, and 30
Population: as for outcome 94
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 4 | 4
Units on a scale
  Month 12: number analyzed (Participants) | 3 | 3
  Month 12 | -0.0 (0.14) | -0.0 (0.14)
  Month 24: number analyzed (Participants) | 3 | 3
  Month 24 | -0.2 (0.16) | -0.2 (0.16)
  Month 30: number analyzed (Participants) | 1 | 1
  Month 30 | -0.3 (NA) — Standard deviation could not be calculated for the single participant. | -0.3 (NA) — Standard deviation could not be calculated for the single participant.

96. Secondary Outcome: Number of Participants According to Response to Each EuroQoL 5 Dimension Youth (EQ-5D-Y) 5 Dimensions at Month 12
Description: EQ-5D-Y is participant completed questionnaire designed to assess impact on health related quality of life in children and adolescents <16 years old. It is comprised of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: 1=no problems, 2=some problems, and 3=extreme problems.
Time Frame: Month 12
Population: Full Analysis Set included all participants who had been enrolled in the study. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 57 | 160 | 217 | 24 | 241
Participants
  Mobility, no problems, Month 12 | 45 | 91 | 136 | 0 | 136
  Mobility, some problems, Month 12 | 12 | 52 | 64 | 0 | 64
  Mobility, extreme problems, Month 12 | 0 | 17 | 17 | 24 | 41
  Self-Care, no problems, Month 12 | 22 | 70 | 92 | 3 | 95
  Self-Care, some problems, Month 12 | 25 | 73 | 98 | 7 | 105
  Self-Care, extreme problems, Month 12 | 10 | 17 | 27 | 14 | 41
  Usual Activities, no problems, Month 12 | 40 | 70 | 110 | 4 | 114
  Usual Activities, some problems, Month 12 | 17 | 74 | 91 | 6 | 97
  Usual Activities, extreme problems, Month 12 | 0 | 16 | 16 | 14 | 30
  Pain/Discomfort, no problems, Month 12 | 36 | 101 | 137 | 17 | 154
  Pain/Discomfort, some problems, Month 12 | 21 | 57 | 78 | 7 | 85
  Pain/Discomfort, extreme problems, Month 12 | 0 | 2 | 2 | 0 | 2
  Anxiety/Depression, no problems, Month 12 | 45 | 110 | 155 | 14 | 169
  Anxiety/Depression, some problems, Month 12 | 8 | 41 | 49 | 9 | 58
  Anxiety/Depression, extreme problems, Month 12 | 4 | 9 | 13 | 1 | 14

97. Secondary Outcome: Number of Participants According to Response to Each EQ-5D-Y 5 Dimensions at Month 24
Description: as for outcome 96
Time Frame: Month 24
Population: as for outcome 96
Measure: Count of Participants; unit: Participants
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 58 | 134 | 192 | 15 | 207
Participants
  Mobility, no problems, Month 24 | 48 | 56 | 104 | 0 | 104
  Mobility, some problems, Month 24 | 10 | 55 | 65 | 0 | 65
  Mobility, extreme problems, Month 24 | 0 | 23 | 23 | 15 | 38
  Self-Care, no problems, Month 24 | 32 | 65 | 97 | 1 | 98
  Self-Care, some problems, Month 24 | 21 | 53 | 74 | 5 | 79
  Self-Care, extreme problems, Month 24 | 5 | 16 | 21 | 9 | 30
  Usual Activities, no problems, Month 24 | 42 | 49 | 91 | 6 | 97
  Usual Activities, some problems, Month 24 | 15 | 60 | 75 | 3 | 78
  Usual Activities, extreme problems, Month 24 | 1 | 25 | 26 | 6 | 32
  Pain/Discomfort, no problems, Month 24 | 38 | 80 | 118 | 12 | 130
  Pain/Discomfort, some problems, Month 24 | 19 | 52 | 71 | 3 | 74
  Pain/Discomfort, extreme problems, Month 24 | 1 | 2 | 3 | 0 | 3
  Anxiety/Depression, no problems, Month 24 | 43 | 91 | 134 | 11 | 145
  Anxiety/Depression, some problems, Month 24 | 14 | 41 | 55 | 3 | 58
  Anxiety/Depression, extreme problems, Month 24 | 1 | 2 | 3 | 1 | 4

98. Secondary Outcome: Number of Participants According to Response to EQ-5D-Y 5 Dimensions at Month 30
Description: as for outcome 96
Time Frame: Month 30
Population: as for outcome 96
Measure: Count of Participants; unit: Participants
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 26 | 78 | 104 | 3 | 107
Participants
  Mobility, no problems, Month 30 | 26 | 34 | 60 | 0 | 60
  Mobility, some problems, Month 30 | 0 | 34 | 34 | 0 | 34
  Mobility, extreme problems, Month 30 | 0 | 10 | 10 | 3 | 13
  Self-Care, no problems, Month 30 | 16 | 45 | 61 | 0 | 61
  Self-Care, some problems, Month 30 | 8 | 23 | 31 | 2 | 33
  Self-Care, extreme problems, Month 30 | 2 | 10 | 12 | 1 | 13
  Usual Activities, no problems, Month 30 | 16 | 28 | 44 | 3 | 47
  Usual Activities, some problems, Month 30 | 10 | 40 | 50 | 0 | 50
  Usual Activities, extreme problems, Month 30 | 0 | 10 | 10 | 0 | 10
  Pain/Discomfort, no problems, Month 30 | 17 | 44 | 61 | 3 | 64
  Pain/Discomfort, some problems, Month 30 | 9 | 30 | 39 | 0 | 39
  Pain/Discomfort, extreme problems, Month 30 | 0 | 4 | 4 | 0 | 4
  Anxiety/Depression, no problems, Month 30 | 18 | 48 | 66 | 1 | 67
  Anxiety/Depression, some problems, Month 30 | 8 | 26 | 34 | 1 | 35
  Anxiety/Depression, extreme problems, Month 30 | 0 | 4 | 4 | 1 | 5

99. Secondary Outcome: Change From Baseline in EQ-5D-Y VAS Assessment at Months 12, 24, and 30
Description: EQ-5D-Y is participant completed questionnaire designed to assess impact on health related quality of life in children and adolescents <16 years old. EQ-VAS recorded the participant's self-rated health on a vertical scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline (Day 1) and Months 12, 24, and 30
Population: Full Analysis Set included all participants who had been enrolled in the study. 'Number of Participants Analyzed' signifies all participants in the Full Analysis Set with age <16 years and contributed data to table, may not have evaluable data for every row. 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 177 | 276 | 32 | 308
Units on a scale
  Month 12: number analyzed (Participants) | 45 | 159 | 204 | 24 | 228
  Month 12 | -1.0 (19.84) | -4.3 (23.02) | -3.5 (22.36) | -5.0 (22.94) | -3.7 (22.37)
  Month 24: number analyzed (Participants) | 43 | 133 | 176 | 15 | 191
  Month 24 | -3.0 (15.08) | -5.6 (21.59) | -5.0 (20.19) | -5.9 (14.59) | -5.1 (19.78)
  Month 30: number analyzed (Participants) | 18 | 77 | 95 | 3 | 98
  Month 30 | -1.0 (12.16) | -6.1 (21.71) | -5.1 (20.30) | 5.0 (5.00) | -4.8 (20.07)

100. Secondary Outcome: Change From Baseline in EQ-5D-Y Index Score at Months 12, 24, and 30
Description: EQ-5D-Y is participant completed questionnaire designed to assess impact on health related quality of life in children and adolescents <=16 years old. It is comprised of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: 1=no problems, 2=some problems, and 3=extreme problems. Participants indicated their health state by choosing the appropriate level from each dimension. The 5 digit health states thus obtained for each dimension were then converted into a single median index value. A health state index score was calculated from individual health profiles using a USA scoring algorithm. Health state index scores generally ranged from -0.109 to 1, where, -0.109= the worst health status, 1= full health. Higher the score the better the better quality of life.
Time Frame: Baseline (Day 1) and Months 12, 24, and 30
Population: as for outcome 99
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 177 | 276 | 32 | 308
Units on a scale
  Month 12: number analyzed (Participants) | 45 | 159 | 276 | 24 | 308
  Month 12 | -0.0 (0.12) | -0.0 (0.16) | -0.0 (0.15) | -0.0 (0.13) | -0.0 (0.15)
  Month 24: number analyzed (Participants) | 43 | 133 | 176 | 15 | 191
  Month 24 | 0.0 (0.13) | -0.1 (0.16) | -0.1 (0.16) | -0.0 (0.12) | -0.1 (0.16)
  Month 30: number analyzed (Participants) | 18 | 77 | 95 | 3 | 98
  Month 30 | 0.0 (0.09) | -0.1 (0.18) | -0.1 (0.17) | 0.0 (0.09) | -0.1 (0.17)

101. Secondary Outcome: Change From Baseline in Healthcare Resource Utilization (HRU) Survey Responses: Visit to Primary Care Physician, Emergency Room and Office Visits at Months 12, 24, and 30
Description: HRU questionnaire is completed by the caregiver and had questions about healthcare resources utilization related to their child's use of healthcare professionals, emergency room visits, and hospitalizations in past 3 months. Change from baseline in mean number of visits to primary care physician, emergency room and office visits is presented in this outcome measure.
Time Frame: Baseline (Day 1) and Months 12, 24, and 30
Population: Full Analysis Set included all participants who had been enrolled in the study. Number of Participants Analyzed' signifies all participants in the Full Analysis Set. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 177 | 276 | 36 | 312
Visits
  To Primary Care Physician at Month 12: number analyzed (Participants) | 80 | 158 | 238 | 30 | 268
  To Primary Care Physician at Month 12 | -0.1 (0.27) | -0.0 (0.41) | -0.0 (0.37) | -0.0 (0.18) | -0.0 (0.36)
  To Primary Care Physician at Month 24: number analyzed (Participants) | 75 | 134 | 209 | 23 | 232
  To Primary Care Physician at Month 24 | 0.0 (0.23) | -0.0 (0.41) | -0.0 (0.35) | 0.1 (0.51) | -0.0 (0.37)
  To Primary Care Physician at Month 30: number analyzed (Participants) | 30 | 76 | 106 | 4 | 110
  To Primary Care Physician at Month 30 | -0.1 (0.43) | 0.0 (0.55) | -0.0 (0.53) | 0.0 (0.00) | -0.0 (0.52)
  To General Practitioner at Month 12: number analyzed (Participants) | 80 | 160 | 240 | 30 | 270
  To General Practitioner at Month 12 | -0.1 (0.45) | -0.0 (0.40) | -0.1 (0.42) | -0.1 (0.35) | -0.1 (0.41)
  To General Practitioner at Month 24: number analyzed (Participants) | 75 | 137 | 212 | 23 | 235
  To General Practitioner at Month 24 | 0.0 (0.57) | -0.1 (0.36) | -0.0 (0.44) | -0.2 (0.52) | -0.1 (0.45)
  To General Practitioner at Month 30: number analyzed (Participants) | 30 | 78 | 108 | 4 | 112
  To General Practitioner at Month 30 | -0.1 (0.40) | -0.1 (0.44) | -0.1 (0.43) | 0.0 (0.00) | -0.1 (0.42)
  To ER Due to Disease at Month 12: number analyzed (Participants) | 80 | 160 | 240 | 30 | 270
  To ER Due to Disease at Month 12 | -0.0 (0.11) | 0.0 (0.27) | -0.0 (0.23) | 0.0 (0.00) | -0.0 (0.22)
  To ER Due to Disease at Month 24: number analyzed (Participants) | 75 | 137 | 276 | 23 | 312
  To ER Due to Disease at Month 24 | -0.0 (0.12) | 0.0 (0.10) | 0.0 (0.10) | 0.0 (0.00) | 0.0 (0.09)
  To ER Due to Disease at Month 30: number analyzed (Participants) | 30 | 78 | 108 | 4 | 112
  To ER Due to Disease at Month 30 | -0.0 (0.18) | -0.0 (0.20) | -0.0 (0.19) | 0.0 (0.00) | -0.0 (0.19)
  Office Visits at Month 12: number analyzed (Participants) | 80 | 160 | 240 | 30 | 270
  Office Visits at Month 12 | -1.6 (7.04) | 0.5 (5.58) | -0.2 (6.18) | -3.4 (11.20) | -0.6 (6.96)
  Office Visits at Month 24: number analyzed (Participants) | 75 | 137 | 212 | 23 | 235
  Office Visits at Month 24 | -0.4 (9.09) | 0.5 (6.44) | 0.2 (7.48) | -6.2 (15.70) | -0.5 (8.78)
  Office Visits at Month 30: number analyzed (Participants) | 30 | 78 | 108 | 4 | 112
  Office Visits at Month 30 | -2.0 (12.84) | -0.2 (7.60) | -0.7 (9.32) | -17.0 (32.67) | -1.3 (11.04)

102. Secondary Outcome: Change From Baseline in HRU Survey Responses: Number of Nights in Hospital Due to Disease/Medication for Disease at Months 12, 24, and 30
Description: HRU questionnaire is completed by the caregiver and had questions about healthcare resources utilization related to number of nights in hospital due to disease/dedication for disease in past 3 months. Change from baseline in mean number of nights in hospital due to disease or medication for disease is presented in this outcome measure.
Time Frame: Baseline (Day 1) and Months 12, 24, and 30
Population: Full Analysis Set included all participants who had been enrolled in the study. 'Number of Participants Analyzed' signifies all participants in the Full Analysis Set and contributed data to the table; however, may not have evaluable data for every row. 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Nights
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 177 | 276 | 36 | 312
Nights
  Month 12: number analyzed (Participants) | 80 | 160 | 276 | 30 | 312
  Month 12 | -0.2 (1.02) | -0.2 (1.82) | -0.2 (1.60) | 0.0 (0.00) | -0.2 (1.51)
  Month 24: number analyzed (Participants) | 75 | 137 | 212 | 23 | 235
  Month 24 | -0.2 (1.06) | -0.2 (1.97) | -0.2 (1.70) | 0.2 (0.83) | -0.2 (1.64)
  Month 30: number analyzed (Participants) | 30 | 78 | 108 | 4 | 112
  Month 30 | 0.0 (0.00) | -0.1 (0.79) | -0.1 (0.67) | 0.0 (0.00) | -0.1 (0.66)

103. Secondary Outcome: Change From Baseline in Out-of-Pocket Money of HRU Survey at Months 12, 24 and 30
Description: Caregivers were asked to estimate out-of-pocket costs related to healthcare resource utilization. The number of out of pocket money was defined as the total spent of the past three months in managing child's Duchenne muscular dystrophy.
Time Frame: Baseline (Day 1) and Months 12, 24, and 30
Population: as for outcome 102
Measure: Mean (Standard Deviation); unit: Chinese Yuan (CYN)
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 177 | 276 | 36 | 312
Chinese Yuan (CYN)
  Month 12: number analyzed (Participants) | 80 | 160 | 276 | 30 | 312
  Month 12 | -2748.1 (6100.61) | 476.0 (10947.21) | -598.7 (9713.33) | 1836.7 (6410.95) | -328.1 (9425.78)
  Month 24: number analyzed (Participants) | 75 | 137 | 212 | 23 | 235
  Month 24 | 352.8 (8484.07) | 777.6 (7630.02) | 627.3 (7925.23) | 2326.1 (6126.93) | 793.6 (7773.09)
  Month 30: number analyzed (Participants) | 30 | 78 | 108 | 4 | 112
  Month 30 | -1794.5 (6772.80) | 1213.6 (6820.65) | 378.0 (6909.59) | -675.0 (4592.29) | 340.4 (6828.66)

104. Secondary Outcome: Change From Baseline in Percent Activity Impairment as Per Work Productivity and Activity Impairment Questionnaire Adapted for Caregiving (WPAI:CG) Caregiver Unchanged at Months 12, 24, and 30
Description: WPAI:CG is a self-reported measure of work productivity and impairment, was completed by caregiver, which had four scores: absenteeism (work time missed); presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment/absenteeism plus presenteeism); and activity impairment. Each score was expressed as a percentage (0-100%) with higher score indicating greater impairment and less productivity.
Time Frame: Baseline (Day 1) and Months 12, 24, and 30
Population: as for outcome 102
Measure: Mean (Standard Deviation); unit: Percentage activity impairment
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 177 | 276 | 36 | 312
Percentage activity impairment
  Month 12: number analyzed (Participants) | 56 | 131 | 187 | 25 | 212
  Month 12 | -6.6 (30.71) | 5.6 (32.08) | 2.0 (32.09) | -6.8 (34.37) | 0.9 (32.41)
  Month 24: number analyzed (Participants) | 54 | 103 | 157 | 19 | 176
  Month 24 | 7.4 (32.22) | 8.8 (34.68) | 8.3 (33.76) | -7.9 (31.02) | 6.6 (33.77)
  Month 30: number analyzed (Participants) | 12 | 55 | 67 | 1 | 68
  Month 30 | -6.7 (31.14) | 13.8 (30.82) | 10.1 (31.65) | 0.0 (NA) — Standard deviation could not be calculated for single participant. | 10.0 (31.43)

105. Secondary Outcome: Change From Baseline in Percent Work Time Missed as Per WPAI: CG Caregiver Unchanged at Month 12
Description: as for outcome 104
Time Frame: Baseline (Day 1) and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage work time missed
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 35 | 58 | 93 | 11 | 104
Percentage work time missed | -6.1 (25.47) | -5.0 (25.17) | -5.5 (25.15) | 3.7 (18.59) | -4.5 (24.63)

106. Secondary Outcome: Change From Baseline in Percent Work Time Missed as Per WPAI: CG Caregiver Unchanged at Month 24
Description: as for outcome 104
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage work time missed
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 33 | 41 | 74 | 11 | 85
Percentage work time missed | 1.1 (24.46) | 0.9 (29.04) | 1.0 (26.91) | -4.4 (23.92) | 0.3 (26.47)

107. Secondary Outcome: Change From Baseline in Percent Work Time Missed as Per WPAI: CG Caregiver Unchanged at Month 30
Description: as for outcome 104
Time Frame: Baseline (Day 1) and Month 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage work time missed
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 9 | 19 | 28 | 1 | 29
Percentage work time missed | -21.5 (26.90) | 2.0 (14.15) | -5.6 (21.73) | 0.0 (NA) — Standard deviation could not be calculated for single participant. | -5.4 (21.36)

108. Secondary Outcome: Change From Baseline in Percent Overall Work Impairment WPAI: CG Caregiver Unchanged at Months 12, 24, and 30
Description: as for outcome 104
Time Frame: Baseline (Day 1) and Months 12, 24, and 30
Population: as for outcome 102
Measure: Mean (Standard Deviation); unit: Percentage work impairment
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 177 | 276 | 36 | 312
Percentage work impairment
  Percent Overall Work Impairment, Month 12: number analyzed (Participants) | 35 | 57 | 92 | 10 | 102
  Percent Overall Work Impairment, Month 12 | -5.2 (26.25) | 2.6 (25.35) | -0.4 (25.83) | -9.3 (36.17) | -1.3 (26.93)
  Percent Overall Work Impairment, Month 24: number analyzed (Participants) | 33 | 40 | 73 | 10 | 83
  Percent Overall Work Impairment, Month 24 | 0.2 (27.83) | 4.8 (26.78) | 2.7 (27.16) | -12.7 (39.72) | 0.9 (29.09)
  Percent Overall Work Impairment, Month 30: number analyzed (Participants) | 9 | 19 | 28 | 1 | 29
  Percent Overall Work Impairment, Month 30 | -11.9 (35.09) | 6.8 (24.29) | 0.8 (28.94) | 30.0 (NA) — Standard deviation could not be calculated for single participant. | 1.8 (28.93)
  Percent impairment while working, Month 12: number analyzed (Participants) | 99 | 58 | 93 | 36 | 103
  Percent impairment while working, Month 12 | -3.7 (19.87) | 4.7 (24.08) | 1.5 (22.84) | -14.0 (33.40) | 0.0 (24.29)
  Percent impairment while working, Month 24: number analyzed (Participants) | 33 | 42 | 75 | 36 | 85
  Percent impairment while working, Month 24 | -1.2 (25.47) | 3.1 (26.82) | 1.2 (26.15) | -15.0 (37.49) | -0.7 (27.94)
  Percent impairment while working, Month 30: number analyzed (Participants) | 9 | 19 | 28 | 1 | 29
  Percent impairment while working, Month 30 | 1.1 (28.48) | 5.3 (25.03) | 3.9 (25.72) | 30.0 (NA) — Standard deviation could not be calculated for single participant. | 4.8 (25.72)

109. Secondary Outcome: Percent Activity Impairment Score as Per WPAI: CG at Months 12, 24, and 30
Description: as for outcome 104
Time Frame: Months 12, 24, and 30
Population: as for outcome 102
Measure: Mean (Standard Deviation); unit: Percentage activity impairment
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 177 | 276 | 36 | 312
Percentage activity impairment
  Month 12: number analyzed (Participants) | 80 | 160 | 240 | 30 | 270
  Month 12 | 30.9 (26.63) | 48.3 (29.02) | 42.5 (29.36) | 61.7 (31.63) | 44.6 (30.17)
  Month 24: number analyzed (Participants) | 75 | 137 | 212 | 23 | 235
  Month 24 | 41.3 (29.38) | 51.8 (27.98) | 48.1 (28.85) | 62.6 (32.78) | 49.5 (29.50)
  Month 30: number analyzed (Participants) | 30 | 78 | 108 | 4 | 112
  Month 30 | 23.7 (23.41) | 56.2 (26.49) | 47.1 (29.45) | 65.0 (31.09) | 47.8 (29.55)

110. Secondary Outcome: Percent Work Time Missed Score as Per WPAI: CG at Month 12
Description: as for outcome 104
Time Frame: Month 12
Population: Full Analysis Set included all participants who had been enrolled in the study. 'Number of Participants Analyzed' signifies all participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage work time missed
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 58 | 89 | 147 | 16 | 163
Percentage work time missed | 6.8 (14.98) | 7.3 (14.11) | 7.1 (14.41) | 21.1 (28.81) | 8.5 (16.78)

111. Secondary Outcome: Percent Work Time Missed Score as Per WPAI: CG at Month 24
Description: as for outcome 104
Time Frame: Month 24
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Percentage work time missed
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 60 | 71 | 131 | 15 | 146
Percentage work time missed | 10.5 (19.70) | 13.0 (23.10) | 11.9 (21.56) | 8.7 (16.50) | 11.5 (21.07)

112. Secondary Outcome: Percent Work Time Missed Score as Per WPAI: CG at Month 30
Description: as for outcome 104
Time Frame: Month 30
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Percentage work time missed
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 27 | 40 | 67 | 3 | 70
Percentage work time missed | 2.9 (6.67) | 13.8 (19.15) | 9.4 (16.21) | 0.0 (0.00) | 9.0 (15.97)

113. Secondary Outcome: Percent Overall Work Impairment Scores as Per WPAI: CG at Months 12, 24, and 30
Description: as for outcome 104
Time Frame: Months 12, 24, and 30
Population: as for outcome 102
Measure: Mean (Standard Deviation); unit: Percentage work impairment
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Total Ambulatory Participants | Non-ambulatory Participants | Total Participants
Number analyzed (Participants) | 99 | 177 | 276 | 36 | 312
Percentage work impairment
  Percent Overall Work Impairment, Month 12: number analyzed (Participants) | 58 | 89 | 147 | 15 | 162
  Percent Overall Work Impairment, Month 12 | 32.0 (25.70) | 45.1 (26.4) | 39.9 (26.60) | 46.6 (29.38) | 40.5 (26.85)
  Percent Overall Work Impairment, Month 24: number analyzed (Participants) | 59 | 70 | 129 | 15 | 144
  Percent Overall Work Impairment, Month 24 | 37.2 (27.64) | 44.3 (27.53) | 41.1 (27.70) | 45.9 (29.86) | 41.6 (27.86)
  Percent Overall Work Impairment, Month 30: number analyzed (Participants) | 27 | 40 | 67 | 3 | 70
  Percent Overall Work Impairment, Month 30 | 23.3 (24.41) | 51.9 (25.52) | 40.4 (28.63) | 56.7 (20.82) | 41.1 (28.42)
  Percent impairment while working, Month 12: number analyzed (Participants) | 59 | 89 | 147 | 15 | 162
  Percent impairment while working, Month 12 | 27.9 (23.90) | 41.3 (25.01) | 36.1 (25.36) | 40.7 (26.58) | 36.5 (25.43)
  Percent impairment while working, Month 24: number analyzed (Participants) | 59 | 71 | 130 | 15 | 145
  Percent impairment while working, Month 24 | 32.5 (24.95) | 37.7 (25.92) | 35.4 (25.52) | 41.3 (28.00) | 36.0 (25.75)
  Percent impairment while working, Month 30: number analyzed (Participants) | 27 | 40 | 67 | 3 | 70
  Percent impairment while working, Month 30 | 21.1 (24.23) | 45.3 (24.60) | 35.5 (27.04) | 56.7 (20.82) | 36.4 (27.03)

ADVERSE EVENTS:
Time Frame: Up to Month 30
Arm/Group | Ambulatory Participants With Age <6 Years | Ambulatory Participants With Age >=6 Years | Non-ambulatory Participants
All-Cause Mortality (participants affected / at risk) | 1/99 | 0/177 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/177 | 0/36
Other Adverse Events (participants affected / at risk) | 84/99 | 136/177 | 20/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ambulatory Participants With Age <6 Years (N=99) | Ambulatory Participants With Age >=6 Years (N=177) | Non-ambulatory Participants (N=36)
Leukocytosis (Blood and lymphatic system disorders) | 19 | 24 | 5
Sinus tachycardia (Cardiac disorders) | 5 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 5 | 2 | 0
Pyrexia (General disorders) | 9 | 7 | 1
Bronchitis (Infections and infestations) | 12 | 4 | 0
COVID-19 (Infections and infestations) | 6 | 22 | 1
Nasopharyngitis (Infections and infestations) | 4 | 10 | 2
Pharyngitis (Infections and infestations) | 5 | 2 | 0
Tonsillitis (Infections and infestations) | 5 | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 74 | 89 | 13
Fall (Injury, poisoning and procedural complications) | 2 | 9 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 10 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT03760029/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT03760029/SAP_001.pdf